#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for a randomized double-blind (sponsor unblind), placebo-controlled, multi-centred phase Ila study to evaluate the safety and efficacy of 13 weeks of once daily oral dosing of the selective androgen receptor modulator (SARM) GSK2881078 in older men and post menopausal women with COPD and muscle weakness, participating in home exercise |
| Compound Number | : | GSK2881078 |
| Effective Date | : | 09-JAN-2020 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 200182 Amendment 3.
- This RAP is intended to describe the safety and efficacy analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables

# RAP Author(s):

# Author PPD Associate Statistician (Respiratory, Biostatistics) Co-Author PPD Principle Biostatistician, (Parexel)

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# RAP Team Reviewers (Method: E-mail)

| Approver | Date |
|---|---|
| PPD | 07-JAN-2020 |
| Clinical Investigation Lead (Discovery Medicine, CPEM) | |
| Medical Monitor, Discovery Medicine Lead, Discovery Medicine, | 07-JAN-2020 |
| CPEM | |
| PPD | |
| Data Quality Lead (Clinical Data Sciences Canada, RD Projects Clinical Platforms & Sciences) | 06-JAN-2020 |
| PPD | 00 1441 0000 |
| Clinical Program Lead (GCSD) | 06-JAN-2020 |
| PPD | |
| Safety Scientist, Safety and Medical Governance Scientist | 06-JAN-2020 |
| PPD | |
| Medical Director, Safety and Medical Governance: | 06-JAN-2020 |
| PPD | |
| Regulatory Affairs (Global Regulatory Affairs) | 06-JAN-2020 |
| PPD | |
| Clinical Pharmacologist (Clinical Pharmacology Modelling and Simulations) | 06-JAN-2020 |
| PPD | |
| Patient Centred Outcomes Lead (Value Evidence and Outcomes) | 08-JAN-2020 |
| PPD | |
| Study Programmer (FPD, Clinical programming) | 08-JAN-2020 |

# **Clinical Statistics and Clinical Programming Line Approvals:**

# (Method: Pharma TMF e-signature)

| Approver | Date |
|-------------------------------------------------|-------------|
| Statistics Director (FPD, Clinical Statistics) | 09-JAN-2020 |
| Programming manager (FPD, Clinical Programming) | 09-JAN-2020 |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | ODUCTIO | ON | 6 |
| 2. | CLIMA | | KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | es to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study ( | Objectives and Endpoints | ٥ |
| | 2.2. | | Design | |
| | 2.4. | | cal Analyses | |
| | ۷.٦. | Otalistic | Sai Analyses | 12 |
| 3. | PLAN | NED AN | ALYSES | 13 |
| • | 3.1. | | nalyses | |
| | | | , | |
| 4. | ANAL | YSIS PO | PULATIONS | 13 |
| | 4.1. | Protoco | ol Deviations | 14 |
| 5. | CON | /ENTION | TIONS FOR DATA ANALYSES AND DATA HANDLING | 15 |
| | 5.1. | | Freatment & Sub-group Display Descriptors | |
| | 5.2. | | e Definitions | |
| | 5.3. | | ntre Studies | |
| | 5.4. | | nation of Covariates, Other Strata and Subgroups | 17 |
| | | 5.4.1. | Covariates and Other Strata | |
| | | 5.4.2. | | |
| | 5.5. | | Comparisons and Multiplicity | 17 |
| | 5.6. | | Considerations for Data Analyses and Data Handling | 47 |
| | | Conver | ntions | 17 |
| 6. | STUD | V DODLI | LATION ANALYSES | 10 |
| 0. | 6.1. | | ew of Planned Study Population Analyses | |
| | 0.1. | Overvie | ew of Flatified Study Fopulation Arialyses | 10 |
| 7. | EFFIC | CACY AN | IALYSES | 20 |
| | 7.1. | Primary | / Efficacy Analyses | 20 |
| | | 7.1.1. Î | | |
| | | 7.1.2. | Endpoint / Variables | <mark>20</mark> |
| | | 7.1.3. | Population of Interest | 20 |
| | | 7.1.4. | Statistical Analyses / Methods | 20 |
| | | | 7.1.4.1. Statistical Methodology Specification | 20 |
| | 7.2. | Second | dary Efficacy Analyses | <mark>22</mark> |
| | | 7.2.1. | Endpoint / Variables | <mark>22</mark> |
| | | 7.2.2. | Summary Measure | <mark>23</mark> |
| | | 7.2.3. | Population of Interest | <mark>24</mark> |
| | | 7.2.4. | Statistical Analyses / Methods | <mark>24</mark> |
| | | | 7.2.4.1. Statistical Methodology Specification | 24 |
| | 7.3. | • | atory Efficacy Analyses | |
| | | 7.3.1. | Endpoint / Variables | |
| | | 7.3.2. | Summary Measure | |
| | | 7.3.3. | Population of Interest | |
| | | 7.3.4. | Statistical Analyses / Methods | |
| | | | 7.3.4.1. Statistical Methodology Specification | 28 |

#### **CONFIDENTIAL**

| | | 7.3.4.2. Other Analyses | 29 |
|---|---|---|---|
| 8. | SAFET<br>8.1. | TY ANALYSESAdverse Events Analyses | |
| | 8.2. | Adverse Events of Special Interest Analyses | |
| | 8.3. | Clinical Laboratory Analyses | |
| | 8.4. | Other Safety Analyses | |
| | 0.4. | Other Salety Analyses | 31 |
| 9. | PHAR | MACOKINETIC ANALYSES | 32 |
| 10. | POPU | LATION PHARMACOKINETIC (POPPK) ANALYSES | 32 |
| 11. | REFE | RENCES | 33 |
| 12. | | NDICES | 34 |
| | 12.1. | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population | 34 |
| | | 12.1.1. Exclusions from Per Protocol Population | |
| | 12.2. | Appendix 2: Schedule of Activities | |
| | 12.2. | 12.2.1. Protocol Defined Schedule of Events | |
| | 12.3. | Appendix 3: Assessment Windows | |
| | 12.5. | 12.3.1. Definitions of Assessment Windows for Analyses | |
| | 12.4. | Appendix 4: Study Phases | |
| | 12.7. | 12.4.1. Study Phases | |
| | | 12.4.2. Study Phases for Concomitant Medication | |
| | 12.5. | Appendix 5: Data Display Standards & Handling Conventions | |
| | 12.5. | 12.5.1. Reporting Process | |
| | | 12.5.2. Reporting Standards | |
| | 12.6. | Appendix 6: Derived and Transformed Data | |
| | 12.0. | 12.6.1. General | |
| | | , | |
| | 10.7 | 12.6.3. Safety | |
| | 12.7. | Appendix 7: Reporting Standards for Missing Data | |
| | | 12.7.1. Premature Withdrawals | |
| | | 12.7.2. Handling of Missing Data | |
| | 40.0 | 12.7.2.1. Handling of Missing and Partial Dates | |
| | 12.8. | Appendix 8: Values of Potential Clinical Importance | |
| | | 12.8.1. Laboratory Values | |
| | | 12.8.2. ECG | |
| | 40.0 | 12.8.3. Vital Signs | 54 |
| | 12.9. | Appendix 9: Model Checking and Diagnostics for Statistical | |
| | 10.10 | Analyses | 55 |
| | 12.10. | Appendix 10: Abbreviations & Trade Marks | |
| | | 12.10.1. Abbreviations | |
| | | 12.10.2. Trademarks | |
| | 12.11. | Appendix 11: List of Data Displays | |
| | | 12.11.1. Data Display Numbering | |
| | | 12.11.2. Mock Example Shell Referencing | <u>5</u> 9 |
| | | 12.11.3. Deliverables | |
| | | 12.11.4. Study Population Tables | |
| | | 12.11.5. Efficacy Tables | |
| | | 12.11.6. Efficacy Figures | 69 |

#### **CONFIDENTIAL**

| 12.11.7. Safety Tables | 70 |
|-----------------------------------------------------------|----|
| 12.11.8. Safety Figures | |
| 12.11.9. Pharmacokinetics Tables | |
| 12.11.10.ICH Listings | |
| 12.11.11.Non-ICH Listings | |
| 12.12. Appendix 12: Example Mock Shells for Data Displays | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol.

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| <ul> <li>An interim analysis for the<br/>assessment of futility is<br/>planned (Section 5.1 in the<br/>protocol).</li> </ul> | Removed all references<br>to the interim analysis | <ul> <li>Decided to cancel the<br/>planned interim analysis,<br/>as per the Note to File<br/>dated 5March2019</li> </ul> |
| A multivariate Bayesian approach using non-informative priors will be employed, data permitting, to further explore the relationships between changes in strength and lean mass and the functional outcomes (ISWT, ESWT,) and to inform decision making. (Section 10.3.3 in the protocol) | Multivariate Bayesian<br>approach will not be<br>planned | Decision making endpoints will be analysed using a univariate Bayesian approach and a decision-making framework prospectively defined for these endpoints. Any multivariate Bayesian analyses will be considered as post-hoc analysis if data warranted. |
| • NA | Analysis of % change from baseline in appendicular, and total lean mass as assessed by Dual-energy X-ray Absorptiometry (DXA) will be planned | To assist clinical team<br>review of the secondary<br>endpoints |
| • NA | Analysis of % change from baseline in Constant Work Rate (CWR) duration from endurance shuttle walking test and peak performance from incremental shuttle | To assist clinical team<br>review of the secondary<br>endpoints |

| Pro | otocol | Reporting & Analy | sis Plan | |
|---|---|---|---|---|
| Sta | tistical Analysis Plan | Statistical Analysi | | ationale for Changes |
| | · | walking test w<br>planned | vill be | Ū |
| • | NA | The responde<br>and analysis be<br>treatment grow<br>(GSK2881078)<br>for COPD Asse<br>Test (CAT) and<br>George Respondance<br>Questionnaire<br>(SGRQ-c) will | petween ups B/ Placebo) sessment nd St iratory e-COPD | To assist clinical team review of the secondary endpoints |
| • | NA | <ul> <li>A Bayesian as<br/>added for the<br/>'times for chair</li> </ul> | endpoint | To assist clinical team review of the secondary endpoints |
| • | Log-transformed leg press<br>strength data will be conducted<br>as supportive analysis of the<br>primary endpoint | <ul> <li>Log-transform<br/>press strength<br/>be analysed of<br/>the model ass<br/>are not met, a<br/>transformation<br/>applicable</li> </ul> | n data will<br>only when<br>sumptions<br>and log-<br>n is | analysed by appropriate methods, therefore transformations of the data prior to analysis will only be done if applicable. |
| • | Log-transformed supportive analysis for all the endpoints in case of violation of assumptions | will be analyse when the mod assumptions a met, and log-transformation applicable | ed only<br>lel<br>are not | Data will only be analysed by appropriate methods, therefore transformations of the data prior to analysis will only be done if applicable. |
| • | Exploratory endpoint: Further exploratory analyses may include changes from baseline in size of inspiratory muscles and/ or other organs. | • Will not analys | sed in this • | There is no data collected |
| • | Exploratory endpoint: Gain further insights into the participants' experience with study treatment and their participation in the trial. | • Will not analys | sed in this • | Exit interview data will be reported separately |
| • | The 'Analysis Population' (AP) is defined as participants in the 'All Participants' population having baseline and at least one post-baseline assessment of the strength, lean mass or functional endpoint (Section | The 'Analysis Population' (defined as point the 'All Papopulation has baseline and one post-baseline and post-basel | AP) is<br>articipants<br>rticipants'<br>aving<br>I at least | The endpoint PROactive scores also added to the definition. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan 10.2 in the protocol). | Statistical Analysis Plan assessment of the lean mass or PROactive scores or any of the functional endpoints. | Rationale for Changes |
| The 'Per Protocol Population' will consist of any AP participants who are compliant with protocol-specific criteria and who do not experience an exacerbation during the treatment phase of the study. Participants with specified protocol deviations and those failing to complete the Week 13 functional assessments will be excluded (Section 10.2 in the protocol). | The 'Per Protocol Population' will consist of any AP participants who are compliant with protocol-specific criteria and who do not experience an exacerbation during the treatment phase of the study. Participants with specified protocol deviations and those failing to complete the Week 13 functional assessments or PROactive scores or lean mass will be excluded. | The endpoint PROactive scores also added to the definition. |

# 2.2. Study Objectives and Endpoints

| Ob | ectives | Endpoints |
|---|---|---|
| Pri | mary Objectives | Primary Endpoints |
| • | Assess the safety and tolerability of approximately 13 weeks of dosing of GSK2881078. | <ul> <li>Safety and tolerability of GSK2881078 as assessed<br/>by clinical monitoring of blood pressure, heart rate,<br/>electrocardiogram (ECG) and laboratory safety data,<br/>as well as reporting of adverse events (AEs)</li> </ul> |
| • | Assess the effect of approximately 13 weeks of dosing of GSK2881078 on leg strength in older men and postmenopausal women with COPD and muscle weakness, participating in home exercise. | % change from baseline and change from baseline in<br>maximum leg press strength following 1 repetition<br>maximum (1- RM) |
| Sec | condary Objectives | Secondary Endpoints |
| • | Assess the effect of approximately 13 weeks of dosing of GSK2881078 on lean soft tissue mass. | <ul> <li>Change from baseline in appendicular, and total lean<br/>mass as assessed by Dual-energy X-ray<br/>Absorptiometry (DXA).</li> </ul> |
| • | Assess the effect of approximately 13 weeks of dosing of GSK2881078 on exercise capacity. | Change from baseline in total Short Physical<br>Performance Battery (SPPB) score and times for<br>chair rise and 4 m gait speed. |
| | | <ul> <li>Change from baseline in Constant Work Rate<br/>(CWR) duration from endurance shuttle walking<br/>test.</li> </ul> |
| | | Change from baseline in peak performance from incremental shuttle walking test. |
| • | Assess the effect of approximately 13 weeks of dosing of | Change from baseline in COPD Assessment Test (CAT). |
| | GSK2881078 on patient reported outcomes, levels of physical activity, activities of daily living and the patient perspective of efficacy. | Change in PROactive endpoints (individual components and total score). |
| | | Change in physical activity measures as assessed via an accelerometer. |
| | | Patient Global Impression of Change. |
| | | Patient Global Rating of Severity. |
| | | Change in St George Respiratory Questionnaire-<br>COPD (SGRQ-c) total score and domains |
| • | Assess the effect of approximately 13 weeks of dosing of | <ul> <li>Change from baseline in forced expiratory volume in<br/>1 second (FEV1)</li> </ul> |
| | GSK2881078 on respiratory function. | <ul> <li>Change from baseline in Sniff nasal inspiratory<br/>pressure (SnIP).</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Characterise the population pharmacokinetic (PK) profile of approximately 13 weeks of dosing of GSK2881078 in older men and post-menopausal women with COPD and muscle weakness. | Model specific PK parameters of GSK2881078 (e.g., oral clearance, oral steady-state volume of distribution). |
| Exploratory Objectives | Endpoints |
| Assess the safety of 13 weeks of dosing of GSK2881078 in older men and postmenopausal women in a subset of up to 15 male and 15 female participants with COPD via magnetic resonance imaging (MRI). | Changes from baseline in hepatic, prostate (males) and cardiac structure and function as assessed via MRI. Further exploratory analyses may include changes from baseline in size of inspiratory muscles and/ or other organs. |
| Conduct semi-structured exit interviews. | Gain further insights into the participants' experience with study treatment and their participation in the trial. |
| Assess the effect of 13 weeks of dosing of GSK2881078 in older men and postmenopausal women on peripheral strength. | <ul> <li>Changes from baseline in handgrip strength.</li> <li>Potentially explore adherence to exercise program (daily physical activity and thrice-weekly strengthening exercises).</li> </ul> |

#### 2.3. Study Design



| Overview of Study Design and Key Features | |
|---|---|
| Interim | No interim analysis is planned for the study (See Note to File dated) |
| Analysis | 5March2019) |

# 2.4. Statistical Analyses

Change from baseline and percent change from baseline in maximum leg press strength following 1- RM will be analyzed separately using mixed models repeated measures (MMRM) models with effects for treatment, day, treatment x day, and baseline strength. Differences in least squares means between the GSK2881078 treated group and placebo treated group will be calculated (i.e.; GSK2881078 - placebo) along with associated 90% CIs. The analysis will be done separately for each gender.

The analyses will be performed using all available data from participants in both the analysis population and the Per Protocol Population. The effects of potential predictors of response including baseline BMI and percent predicted FEV1 will be explored.

Additionally, a Bayesian approach using a non-informative prior will be conducted to estimate the posterior distribution and to estimate the probability that the true treatment difference of % change from baseline strength at week 13 (Day90) is  $\geq$  9%. Additional threshold values and timepoints will also be presented for all decision-making endpoints including other key secondary endpoints.

Model and distributional assumptions underlying each analysis will be assessed and the details can be found at Appendix 9.

Safety data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. No formal statistical comparisons will be made for the safety data.

Sample size estimations and explorations into sample size sensitivity are given in Section 10.1 of the protocol.

#### 3. PLANNED ANALYSES

# 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | <ul> <li>All participants who were screened for eligibility<br/>and allocated a subject number.</li> </ul> | Screened subjects |
| Enrolled | <ul> <li>All participants who passed screening and entered the study.</li> <li>Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Study Population |
| All Participants | <ul> <li>The 'All Participants Population' is defined as all randomized participants who receive at least one dose of study medication.</li> <li>This population will be based on the treatment the participant was randomized to.</li> </ul> | Study Population |
| Safety | <ul> <li>The 'Safety Population' is defined as all randomized participants who receive at least one dose of study medication.</li> <li>This population will be based on the treatment the participant received.</li> </ul> | Safety |
| Analysis (AP) | <ul> <li>The 'Analysis Population' (AP) is defined as participants in the 'All Participants' population having baseline and at least one post-baseline assessment of the lean mass or PROactive scores or any of the functional endpoints.</li> <li>This population will be based on the treatment the participant was randomized to. The functional endpoints include leg press strength, peak performance from Incremental shuttle walking test, Constant Work Rate (CWR) duration from endurance shuttle walking test, total SPPB score and handgrip strength.</li> </ul> | • Efficacy |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Per Protocol | The 'Per Protocol Population' will consist of any AP participants who are compliant with protocol-specific criteria and who do not experience an exacerbation during the treatment phase of the study. Participants with specified protocol deviations and those failing to complete any of the Week 13 functional assessments or PROactive scores or lean mass will be excluded. This population will be based on the treatment the participant was randomized to. Further details will be given in <a href="Section 12.1.1">Section 12.1.1</a> . | Efficacy (Strength,<br>SGRQ, PROactive<br>Constant Work<br>Rate (CWR)<br>duration from<br>endurance shuttle<br>walking test and<br>time for repeated<br>chair rise) |
| Pharmacokinetic (PK) | The 'PK Population' is defined as participants in the<br>'All Participants' population for whom a PK sample was<br>obtained and analysed for GSK2881078. | • PK |

<sup>1.</sup> Refer to Appendix 11: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to <u>Appendix 1</u>: Protocol Deviation Management and Definitions for Per Protocol Population).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the 'Protocol Deviation Specification-version 6.0 dated 28 Nov 2019

- Obata will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset. It will not be possible to identify whether subjects received a different treatment to the one they were randomised to until post unblinding, hence this protocol deviation will be identified after unblinding the database.
- A blinded data review meetings (BDRM) will be handled before the final database release (DBR)
- This dataset will be the basis for the summaries and listings of protocol deviations.

A listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

The analysis and summary will be separately analysed by gender. All graphical displays will present results for males and females on separate pages. Sex will be either a subtitle or subheading ("by" variable) on these displays.

For each efficacy analysis table, the results for female will displayed first and then repeated for male; for other tables, the summary will be presented in the order of female and male. Listings will be sorted by gender.

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | Treatment Group Data Displays for Reporting | | |
| Code | Description | Description Order i | |
| Α | PTM GSK2881078 1.0mg | Placebo | 1 - Female |
| В | GSK2881078 1.0 mg | GSK2881078 1.0 mg | 2- Female |
| С | PTM GSK2881078 2.0mg | Placebo | 1 - Male |
| D | GSK2881078 2.0 mg | GSK2881078 2.0 mg | 2- Male |

Treatment comparisons will be displayed as follows using the descriptors as specified and separated by gender:

Female: GSK2881078 1.0 mg vs Placebo Male: GSK2881078 2.0 mg vs Placebo

#### 5.2. Baseline Definitions

| Parameter | Study A | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| | Screening | Day -9 | Day 1 (Pre-Dose) | |
| Efficacy | | | | |
| Leg Strength | Χ | | Х | whichever is latest* |
| Incremental Shuttle Walk Test | | Х | X | whichever is higher |
| Endurance Shuttle Walk Test | | | Х | Day 1 |
| Dual-energy X-ray Absorptiometry (DXA) | | | Х | Day 1 |
| Short Physical Performance<br>Battery (SPPB) | Х | | Х | whichever is latest* |
| COPD Assessment Test (CAT) | | | Х | Day 1 |
| Patient Global Rating of Severity (PGRS) | | | Х | Day 1 |
| St George Respiratory | | | Х | Day 1 |

| Parameter | Study As | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| | Screening | Day -9 | Day 1 (Pre-Dose) | |
| Questionnaire COPD (SGRQ-c) | | | | |
| PROactive Physical Activity | Х | Χ | | See detail below** |
| Spirometry | X | | X | whichever is latest* |
| Sniff Nasal Inspiratory Pressure (SnIP) | Х | | X | whichever is latest* |
| Safety | | | | |
| Vital Signs | Х | | X | whichever is latest* |
| 12-lead ECG | Х | | X | whichever is latest* |
| Haematology | Х | | X | whichever is latest* |
| Clinical Chemistry | Х | | X | whichever is latest* |
| Urinalysis | Х | | X | whichever is latest* |
| hsCRP, Fibrinogen | | | X | Day 1 |
| Lipid panel | Х | | X | whichever is latest* |
| PSA | Х | | X | whichever is latest* |
| HbA1c | X | | | screening |
| Exploratory | | | | |
| Cardiac and liver MRI | | | X | Day 1 |
| Handgrip strength | X | | X | whichever is latest* |
| Reproductive Tissue Biomarkers | | | X | Day 1 |
| Bone Biomarkers | | | X | Day 1 |
| ***Exploratory Biomarkers | | | X | Day 1 |
| ***Monitored home exercise program | | Х | Х | whichever is latest* |

<sup>\*</sup>Baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

<sup>\*\*</sup>Baseline will be the average of the data collected from the 7-day period after Day -9 device dispense.

<sup>\*\*\*</sup>Exploratory Biomarkers and home exercise program will be analysed separately and will not be reported as part of this study Statistical Analysis Complete reporting.

#### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site. There is no analysis planned by center/investigative site.

#### 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates which will be used in descriptive summaries and statistical analyses., including the primary analysis are described in the table below. Additional covariates percent predicted FEV1 and baseline BMI will be explored as a sensitivity analysis for the primary endpoint of the leg press strength only.

| Category Details | |
|---|---|
| Covariates | Treatment, Day, Treatment x Day and Baseline |
| Exploratory covariates | Percent Predicted FEV1 and Baseline BMI |

#### 5.4.2. Examination of Subgroups

There is no subgroup analysis planned for this RAP, however, males and females will be analysed separately since they have a different dose level.

## 5.5. Multiple Comparisons and Multiplicity

The primary comparison of interests is the change from baseline and percent change from baseline in maximum leg press strength following 1 repetition maximum (1- RM). The key endpoint used for decision making purpose will be the percent change from baseline in maximum leg press strength. This analysis will be conducted separately for each gender and the two analyses will be considered co-primary (i.e. both must be considered a success for the study to be successful), therefore no multiplicity adjustment is required. There will be no multiplicity adjustments for multiple endpoints or multiple timepoints or multiple treatment comparisons. Analyses of other efficacy endpoints will not be subject to any multiplicity adjustment.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|-----------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be mainly based on the All Participants population unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in <u>Appendix 11</u>: List of Data Displays.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data Displa | y's Generated |
|---|---|---|
| | Table | Listing |
| Randomisation | | • |
| Randomisation | | Y [1] |
| Subject Disposition | | |
| Subjects Enrolled by Country and Site ID [6] | Υ | Y |
| History of Rescreened Subjects [2] | | Y |
| Reasons for Screen Failure [2] | Υ | Υ |
| Subjects for Whom the Treatment Blind was Broken | | Y |
| Subject Disposition | Υ | Y |
| Study Visit Dates | | Y |
| Populations Analysed | | |
| Study Populations [2] | Y | Y |
| Protocol deviations | | |
| Important Protocol Deviations | Υ | Y |
| Deviations leading to exclusion from PP | Υ | Y |
| Inclusion and Exclusion Criteria Deviations | | Υ |
| Demography | | |
| Demographic Characteristics [3] | Υ | Y |
| Summary of Age Ranges [6] | Υ | |
| Race & Racial Combinations [4] | Υ | Y |
| Disease Staging | | Υ |
| Medical Conditions, Concomitant Medications | | |
| Medical Conditions (Current and Past) | Υ | Υ |

| Exacerbation History | | Y |
|---|---|---|
| Alcohol History | | Y |
| History of Tobacco Use | | Y |
| Change of Smoking Status During the Study | | Y |
| Concomitant Medications | Υ | Y |
| HIV, Hepatitis B and C screening (Hepatitis C viral RNA PCR if Hepatitis C screening is positive) | | Y |
| Other | | |
| IP Compliance [5] | Y | Y |

#### NOTES:

- Y = Display Generated, T = Tables, L = Listings, IP = Investigational Product
- 1. One listing of subjects randomised but not treated.
- 2. Screened population.
- 3. Age, sex, age group, ethnicity, race, weight, height, body surface area, percent predicted FEV1 and BMI (kg/m^2) needs to be summarized.
- 4. The five-high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high-level categories which exist in the data. A by-subject listing of race will also be produced.
- 5. Dispensation information (dates, number of tablets dispensed, returned, taken and lost, compliance percentage, duration of treatment and treatment cumulative dose also will be included).
- 6. Enrolled population

#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

#### 7.1.1. Summary Measure

The adjusted mean treatment difference for change and percent change from baseline in maximum leg press strength will be presented at Days 28, 56 and 90.

#### 7.1.2. Endpoint / Variables

The primary endpoints are change from baseline and percent change from baseline in maximum leg press strength following 1 repetition maximum (1- RM). The key endpoint used for decision making purpose will be the percent change from baseline in maximum leg press strength.

#### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Analysis population. A supportive efficacy analyses will be based on the Per Protocol population.

#### 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in <u>Appendix 11</u>: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in <u>Section 7.1.1</u> will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.1.4.1. Statistical Methodology Specification

#### **Endpoints / Variables**

% change from baseline and change from baseline in maximum leg press strength (Kg) following 1 repetition maximum (1- RM) at Days 28, 56 and 90.

#### **Model Specification**

- Change from baseline and percent change from baseline strength will be analyzed separately using mixed models repeated measures (MMRM) adjusted for treatment, day, treatment x day, and baseline strength, with day as the repeated factor.
- Data falling into the analysis windows for day 28, day 56 and day 90 will be included in the model
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- In the event that this model fails to converge, the model will be re-fitted with other covariance structures such as compound symmetry and one which gives the least Akaike's Information Criteria (AIC) from the fitted model will be used as the covariance structure.
- The analysis will be conducted separately by gender

• If there are any departures from the distributional assumptions for change or percentage change from baseline, the change of log-transformed data at post- baseline from log baseline will be the response variable, adjusted for treatment, log-transformed baseline strength, day and the interaction of treatment and day, with day as the repeated factor. The sensitivity analysis for the change from baseline and percentage change from baseline are the same.

#### **Model Checking & Diagnostics**

Refer to <u>Appendix 9</u>: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- For change and percent change from baseline, adjusted means, corresponding standard error
  of means (SEs) and 90% confidence intervals will be presented for each treatment by day,
  together with estimated treatment differences (GSK2881078 Placebo) and the corresponding
  90% confidence intervals and p-value by day for both Analysis and Per Protocol population.
- A line plot of the adjusted mean of change (and percentage change) from baseline as well as the 90% confidence interval over time (day) for each treatment from the MMRM model will be provided for the analysis population.

#### Log-transformed data results presentation

- The estimated coefficients of the MMRM model will be transformed back (exponential transform).
- For each treatment, adjusted ratio of the post baseline value to the baseline value and corresponding 90% confidence intervals will be presented by day.
- The adjusted treatment ratio of the ratio (postbaseline value/baseline value) between the two
  treatments with the corresponding 90% confidence interval be presented by day.
- The plot of adjusted ratio of the post baseline value to the baseline value and its 90% confidence interval over time (day) for each treatment arm will be presented for the analysis population

# **Supportive Statistical Analysis - Bayesian**

- % change from baseline in maximum leg press strength following 1 repetition maximum (1-RM) at Days 28, 56 and 90 will be estimated by Bayesian analysis and separately by gender.
- The posterior probability of treatment difference greater than 4% points, less than 9% points and greater than or equal to 9% points for each visit separately by gender.

#### **Model Specification**

- Create indicator variables for the categorical effect: Treatment (GSK2881078 vs. Placebo) and Day (day28, day56 and day90).
  - For treatment, if treatment=placebo, then drug=0; if treatment=GSK2881078, then drug=1;
- Construct a linear model for each day(visit) in order to model within-subject observation covariance structures by multivariate normal (MVN) distribution in the MCMC procedure. For subject i on treatment j at Day k, the model can be written as:
  - PCHijk= $\beta$ 0 +  $\beta$ 1 drug +  $\beta$ 2 baseline +  $\beta$ d Dayk +  $\beta$ dk drug\* Dayk + $\epsilon$ ijk  $\epsilon$ ijk

- PROC MCMC from the design matrix. The last element, Day3, is excluded by setting it to 0 in the PARMS statement.
- (β1+ βd1), (β1+ βd2), are the estimated treatment differences (GSK2881078 vs. Placebo) at Day 28, Day 56 respectively. β1 is the estimated treatment difference (GSK2881078 vs. placebo) at Day 90
- Reformat the input data in the way that all repeated measurements from a subject are in one row
- Set seed=123456 with the simulation size of 500000, 5000 burn-in iterations. The simulation size and number of burn-in iterations could be updated during the convergence check.
- The non-informative priors (normal (0, var=1e6)) will be used for the regression parameters
- The 3-dimension inverse wishart scale matrix will be used as the prior of the covariance matrix. The degrees of freedom will be 3 and the positive definite scale matrix will be an identity matrix.
- Multivariate normal (MVN) distribution will be specified to model all repeated measurements
- Count the proportion at Day90 where β<sub>1</sub> greater than 4% points, less than 9% points and greater or equal to 9% points respectively from the posterior probability distribution simulation.
- Similarly, Count the proportion at Day28 and Day56 where  $(\beta_1 + \beta_{d1})$ ,  $(\beta_1 + \beta_{d2})$  are separately greater than 4% points, less than 9% points and greater or equal to 9% points respectively from the posterior probability distribution.
- For calculating the posterior adjusted least square mean and corresponding difference, use the coefficient of L-matrix of the covariates from the MMRM analysis mentioned in <u>Section</u> 7.1.4.1

#### **Model Checking & Diagnostics**

Refer to <u>Appendix 9</u>: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- n, posterior adjusted least square mean and 90% highest posterior density (HPD) interval, the
  adjusted treatment difference and its 90% HPD credible interval and standard deviation for the
  posterior adjusted least square mean and difference.
- The treatment difference (GSK2881078 Placebo) for the percentage change from baseline at each visit (Day 28, Day 56 and Day 90) > 4 percentage points, <9 percentage points and ≥ 9 percentage points will be reported based upon the simulation results from the posterior probability model.

# 7.2. Secondary Efficacy Analyses

# 7.2.1. Endpoint / Variables

The secondary endpoints are:

- Change and % change from baseline in appendicular, and total lean mass as assessed by Dual-energy X-ray Absorptiometry (DXA).
- Change from baseline in total Short Physical Performance Battery (SPPB) score, times for chair rise and 4 m gait speed.

- Change and % change from baseline in Constant Work Rate (CWR) duration from endurance shuttle walking test.
- Change and % change from baseline in peak performance from incremental shuttle walking test.
- Change in PROactive endpoints (individual components (difficulty and amount score) and total score).
- Change from baseline in COPD Assessment Test (CAT).
- Responder of COPD Assessment Test (CAT).
- Change in St George Respiratory Questionnaire (SGRQ) total score and domain scores derived from SGRQ-c raw score.
- Responder of St George Respiratory Questionnaire (SGRQ) defined by the total score.
- Change from baseline in forced expiratory volume in 1 second (FEV1).
- Patient Global Impression of Change (PGIC).
- Patient Global Rating of Severity (PGRS).
- Change from baseline in Sniff nasal inspiratory pressure (SnIP).
- Change in physical activity measures as assessed via an accelerometer.

#### 7.2.2. Summary Measure

The adjusted mean treatment differences (GSK2881078 – Placebo) for the following endpoints will be presented:

- Change and % change from baseline in appendicular, and total lean mass as assessed by Dual-energy X-ray Absorptiometry (DXA) at Days 28, 56 and 90.
- Change from baseline in total Short Physical Performance Battery (SPPB) score, times for chair rise and 4 m gait speed at Days 28, 56 and 90.
- Change and % change from baseline in Constant Work Rate (CWR) duration from endurance shuttle walking test at Day 90.
- Change and % change from baseline in peak performance from incremental shuttle walking test at Day 90.
- Change from baseline in PROactive endpoints at Days 56 and 90. (individual components and total score).
- Change from baseline in COPD Assessment Test (CAT) score at Days 56 and 90.
- Change from baseline in St George Respiratory Questionnaire (SGRQ) total score and domain scores derived from SGRQ-c raw scores at Days 90.

The responder analysis between GSK2881078 and Placebo (GSK2881078/ Placebo) for the following endpoints will be explored

- Odds ratio between treatment groups for the COPD Assessment Test (CAT) responder at Days 56 and 90.
- Odds ratio between treatment groups for the St George Respiratory Questionnaire (SGRQ) responder defined by the total score derived from SGRQ-c raw scores at Days 90.

The descriptive summaries will be reported for the following endpoints

Change from baseline in forced expiratory volume in 1 second (FEV1).

- Frequency and percentages of Patient Global Impression of Change (PGIC) responses.
- Frequency and percentages of Patient Global Rating of Severity (PGRS) responses.
- Change from baseline in Sniff nasal inspiratory pressure (SnIP).
- Change in physical activity measures as assessed via an accelerometer.

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Analysis Population. The decision-making endpoints PROactive endpoint, SGRQ, SPPB (time for repeated chair rise endpoint) and constant work rate (CWR) duration from endurance shuttle walking test will be also analysed based on the Per Protocol population.

#### 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in <u>Appendix 11</u>: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in <u>Section 7.2.1</u> will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.4.1. Statistical Methodology Specification

#### Secondary Efficacy Endpoint / Variables – Multiple Post-baseline Visit

- Change and % change from baseline in appendicular, and total lean mass as assessed by Dual-energy X-ray Absorptiometry (DXA) at Days 28, 56 and 90.
- Change from baseline in total Short Physical Performance Battery (SPPB) score, \*\*time for repeated chair rise and 4 m gait speed at Days 28, 56 and 90.
- Change from baseline (Day 1) in \*PROactive endpoints (individual components (difficulty and amount score) and \*\*total score) at Days 56 and 90.
- Change from baseline in COPD Assessment Test (CAT) score at Days 56 and 90.
- \*A physical activity monitor will be worn for 7 days after the Day -9 visit (Day 1), for 7 days after the Day 56 visit (Day 56), and for 7 days following the day 80 visit (Day 90).
- \*\*Bayesian analysis will be performed only for the endpoints change from baseline of PROactive total scores and change from baseline in the time for repeated chair rise. The posterior probability of treatment difference greater than 3 points and less than 6 points for PROactive total scores and greater than 1.3 seconds and less than 1.7 seconds for time for repeated chair rise will be estimated for each visit separately by gender.

#### **Model Specification**

- Treatment difference (GSK2881078 placebo) at each visit on change from baseline or
  percentage change from baseline (as appropriate) will be analysed using mixed models
  repeated measures (MMRM) models as what was described for the primary efficacy endpoint
  in <u>Section 7.1.4.1</u>. The analyses will be based on the analysis population for all endpoints
  additionally the endpoints PROactive and SPPB will be analysed for per-protocol population as
  well.
- If there are any departures from the distributional assumptions for change or percentage change from baseline, the change of log-transformed data at post- baseline from log baseline will be the response variable, adjusted for treatment, log-transformed baseline value, day and

- the interaction of treatment and day, with day as the repeated factor.
- A Bayesian approach will also be employed for the change from baseline in PROactive weekly total score and time for repeated chair rise to estimate the treatment difference in the change from baseline for analysis population, following the similar procedures described in <u>Section 7.1.4.1</u>. for the primary efficacy endpoint analysis. For calculating the posterior adjusted least square mean and corresponding difference, use the coefficient of L-matrix of the covariates from the corresponding frequentist MMRM analysis.

#### **Model Checking & Diagnostics**

Refer to <u>Appendix 9</u>: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- For change and percent change from baseline, adjusted means and corresponding standard error of means (SEs) and 90% confidence intervals will be presented for each treatment by gender and then by time, together with estimated treatment differences (GSK2881078 – Placebo) and the corresponding 90% confidence intervals for MMRM estimation.
- In case of the violation of assumptions in MMRM analysis, adjusted mean for ratio to baseline and 90% confidence intervals will be presented for each treatment by gender and then by time, together with adjusted treatment ratio of the ratio (postbaseline value/baseline value) between the two treatments with the corresponding 90% confidence interval be presented by day.
- A line plot of the adjusted mean change from baseline or percentage change from baseline (as appropriate) as well as 90% confidence intervals over time (day) for each treatment by gender from the MMRM model will be provided for the analysis population. In case of violation of assumption in MMRM analysis, the adjusted mean for ratio to baseline and corresponding 90% confidence interval will be plotted.
- For the Bayesian analysis, n, posterior adjusted least square mean and 90% highest posterior density (HPD) interval, the adjusted treatment difference and its 90% HPD credible interval and standard deviation for the posterior adjusted least square mean and difference will be reported along with the estimated probabilities.
- For the Bayesian analysis for PROactive weekly total score, the probability of treatment difference (GSK2881078-placebo) greater than 3 points and less than 6 points will be estimated through the simulations of the posterior probability distribution. Similarly, for the Bayesian analysis for time for repeated chair rise, the probability of treatment difference (GSK2881078-placebo) greater than 1.3 seconds and less than 1.7 seconds will be estimated through the simulations of the posterior probability distribution.

# Secondary Efficacy Endpoint / Variables – Categorical Variable

- Odds ratio of COPD Assessment Test (CAT) responder at Days 56 and 90.
- Odds ratio of St George Respiratory Questionnaire (SGRQ) responder derived by the total score at Days 90.

#### **Model Results Presentation**

 The number of responders, odds ratio and associated 90% exact confidence intervals between treatment groups (GSK2881078 vs. placebo) will be reported for CAT and SGRQ responder analysis by gender.

#### Secondary Efficacy Endpoint / Variables - Single Post-baseline Visit

- Change and % change from baseline in Constant Work Rate (CWR) duration\* from endurance shuttle walking test at Day 90.
- Change and % change from baseline in peak performance from incremental shuttle walking test at Day 90.
- Change from baseline in St George Respiratory Questionnaire (SGRQ) total score\* and domain scores derived from SGRQ-c raw scores at Days 90.

\*Bayesian analysis will be performed only for the endpoints change from baseline of Constant Work Rate (CWR) duration and change from baseline of SGRQ total score. The posterior probability of treatment difference greater than 36 seconds and less than 48 seconds for Constant Work Rate (CWR) duration and greater than 2 points and less than 4 points SGRQ total score will be estimated.

#### **Model Specification**

- Treatment difference (GSK2881078 placebo) in the change from baseline and percentage
  change from baseline at Day 90 will be analysed using ANCOVA where baseline and
  treatment will be included as the independent variables in the model. Each gender will be
  analysed separately. The analyses will be based on the analysis population for the endpoints
  CWR duration, peak performance from incremental shuttle walking test and SGRQ total score
  additionally the endpoints CWR duration and SGRQ total score will be analysed for perprotocol population as well.
- If there are any departures from the distributional assumptions, the change of log-transformed data at post- baseline from log baseline will be the response variable, adjusted for treatment, and log-transformed baseline value.
- A Bayesian approach will also be conducted to estimate the treatment difference in the change from baseline at Day 90 for CWR duration and change from baseline SGRQ total score for the analysis population, following the similar procedures described in <u>Section 7.1.4.1</u>. for the primary efficacy endpoint analysis with the model being constructed as below:
- Create indicator variables for the categorical effect: Treatment (GSK2881078 vs. Placebo).
   For treatment, if treatment=placebo, then drug=0; if treatment=GSK2881078, then drug=1;
- For subject i on treatment j, the model can be written as:

$$CH_{ij}=\beta_0 + \beta_1 drug + \beta_2 base + +\epsilon_{ij}$$

where CH refers to the change from baseline at Day 90; base means baseline assessment; drug=0 when treatment is placebo and drug=1 for GSK2881078 treatment;  $\epsilon_{ij} \sim N(0, \sigma^2)$ ;  $\beta_1$  is the estimated treatment difference (GSK2881078 vs. placebo) at Day 90;

- Set seed=123456 with the simulation size of 200000 and 5000 burn-in iterations; the sample size and the number of burn-in iterations could be updated during the convergence check.
- The non-informative priors (normal (0, var=1e6)) will be used for the regression parameters  $\beta_0$ ,  $\beta_1$ , and  $\beta_2$  and the prior for variance  $\sigma^2$  will be the inverse gamma (0.01, scale=0.01)
- For calculating the posterior adjusted least square mean and corresponding difference, use the coefficient of L-matrix of the covariates from the corresponding ANCOVA analysis

#### Model Checking & Diagnostics

• Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- For change and percent change from baseline, adjusted means and corresponding standard error of means (SEs) and 90% confidence intervals will be presented for each treatment at Day 90, together with estimated treatment differences (GSK2881078 – Placebo) and the corresponding 90% confidence intervals through ANCOVA model.
- In case of the violation of assumptions in ANCOVA analysis, adjusted mean for ratio to baseline and 90% confidence intervals will be presented for each treatment by gender, together with adjusted treatment ratio of the ratio (postbaseline value/baseline value) between the two treatments with the corresponding 90% confidence interval be presented.
- For the Bayesian analysis, n, posterior adjusted least square mean and 90% highest posterior density (HPD) interval, the adjusted treatment difference and its 90% HPD credible interval and standard deviation for the posterior adjusted least square mean and difference will be reported along with the estimated probabilities.
- For the Bayesian analysis for CWR duration, the probability of treatment difference (GSK2881078-placebo) greater than 36 seconds and less than 48 seconds will be estimated through the simulations of the posterior probability distribution. Similarly, for the Bayesian analysis for SGRQ total score, the probability of treatment difference (GSK2881078-placebo) greater than 2 points and less than 4 points will be estimated through the simulations of the posterior probability distribution.

#### Secondary Efficacy Endpoint / Variables – Descriptive Summary

- Forced expiratory volume in 1 second (FEV1) at Days 1, 56 and 90.
- Patient Global Impression of Change (PGIC) at Days 14, 28, 56 and 90.
- Patient Global Rating of Severity (PGRS) at Days 1 and 90.
- Sniff nasal inspiratory pressure (SnIP) at Days 1, 56 and 90.
- Physical activity measures as assessed via an accelerometer at Days 1, 56 and 80.

#### **Summary Results Presentation**

Baseline, each postbaseline visit and change from baseline, will be descriptively summarized by treatment group for endpoints: weekly average steps, vector magnitude unit/wear time and moderate/vigorous activity duration measures via an accelerometer. The number of subjects with the eligible days i.e. wear duration more than 8 hours for at least 4 days, the average eligible days for those subjects and average wear duration (minutes) during the eligible days will be summarized.

Baseline, each postbaseline visit and change from baseline, will be descriptively summarized by treatment group for original FEV1 (L) and percentage predicted FEV1 and maximum SnIP.

In addition, a box plot will be prepared for the change from baseline for FEV1 and SnIP at the post-baseline visits.

For the categorical endpoints, PGRS and PGIC, the count and percentage will be summarized by category and treatment for each visit separately by gender.

## 7.3. Exploratory Efficacy Analyses

#### 7.3.1. Endpoint / Variables

The exploratory endpoints that will be analysed are:

Changes from baseline in handgrip strength.

#### 7.3.2. Summary Measure

Descriptive summary of baseline assessments, post-baseline assessments and change from baseline for handgrip strength.

Changes from baseline in size of inspiratory muscles and/or other organs will not be analyzed in this report because there is no data collected. In addition, exit interview data will be reported separately, thus the analysis of the endpoint 'Gain further insights into the participants' experience with study treatment and their participation in the trial' will not be performed in this RAP. The adherence to the exercise program (daily physical activity and thrice-weekly strengthening exercises) will not be explored in this RAP.

#### 7.3.3. Population of Interest

The exploratory efficacy analyses will be based on the Analysis population, unless otherwise specified.

#### 7.3.4. Statistical Analyses / Methods

Details of the planned displays are provided in <u>Appendix 11</u>: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in <u>Section 7.2.1</u> will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.3.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Changes from baseline in handgrip strength.

#### **Summary Results Presentation**

The handgrip strength of left hand and right hand will be separately summarized for baseline,
 Day 90 and change from baseline at Day 90 by treatment for each gender separately

#### 7.3.4.2. Other Analyses

- An exploratory analysis will be performed on the analysis population to identify how the change from baseline of PROactive total and domain scores changes over the responses of PGIC questionnaire. This relationship between PGIC levels and change from baseline in PROactive total and domains scores will be explored by a descriptive summary table for the visits Day 56 and 90. This comparison will be by gender (males, females and overall (male + female)) and not with respect to treatment. Along with the seven levels of PGIC, the pooled categories "Much worse and Worse" and "Better and Much Better" will also be summarized.
- A sensitivity analysis has to be performed to identify the influence of center PPD on the primary analysis. The primary analysis of percentage change from baseline for leg press has to perform by removing the subjects recruited from the center PPD for the analysis population. This is the analysis supporting the SPOOS ((Significant Payments of Other Sorts) impact analysis.

#### Plots to be generated in R-shiny App

Shiny is an open R package from RStudio, which provides a web application framework to create interactive web applications (visualization) called "Shiny apps". Shiny combines the computational power of R with the interactivity of the modern web. Shiny web apps can be deployed locally or on the web through tools such as RStudio Connect.

The below mentioned plots will be generated in the R-shiny app at SAC. These displays will then be sent for clinical review. From the generated plots only the clinically important ones will be identified and added to the CSR and will be considered post hoc analyses. These plots will be generated for the analysis population.

- Absolute, Change and percent change from baseline in the leg press strength and change from baseline in constant work rate (CWR) duration from endurance shuttle walking test and peak performance from incremental shuttle walking test versus baseline SPPB categories will be plotted (box-plot) by treatment group for each gender separately. The box-plots for both the treatment groups will be presented in one plot for one gender; then repeat for the other gender.
- The relationship between absolute, change and percent change from baseline at Day 90 in the leg press strength, change from baseline in constant work rate (CWR) duration from endurance shuttle walking test at Day 90 and peak performance from incremental shuttle walking test at Day 90 versus baseline PROactive scores for all the domains score as well as the baseline average daily steps via an accelerometer will be explored by the scattered plots by treatment group for each gender. Baseline scores will be the x-axis and absolute or change from baseline or percent from baseline at Day 90 in the leg press strength and shuttle walk tests separately will be the y-axis
- Mean absolute, change from baseline and percentage change from baseline in leg press strength, change from baseline in appendicular and total lean mass, constant work rate (CWR) duration from endurance shuttle walking test, peak performance from incremental shuttle walking test, total SPPB score, hand grip, SGRQ (all domains) and PROactive (all domains) will be plotted by treatment group for each gender, where descriptive mean for absolute, change from baseline and percentage change from baseline for the respective endpoints will be the Y-axis in each plot and X-axis will be the visits.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the safety population and actual treatment group, unless otherwise specified. Data for male and female subjects will be analysed separately.

# 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The AE text recorded in the eCRF will be coded using the Medical Dictionary for Regulatory Activities (MedDRA version 22.0) and will be reported using the primary System Organ Class (SOC) and Preferred Term (PT). Results will be displayed irrespective of treatment phase in the order of decreasing frequency, both across SOC and within SOC. The details of the planned displays are provided in <a href="Appendix 11">Appendix 11</a>: List of Data Displays.

For those displays with maximum intensity, if AEs are reported more than once by a subject, the most severe intensity will be included. An adverse event will be considered as a common adverse event if it occurs in more than one patient in either gender.

#### 8.2. Adverse Events of Special Interest Analyses

The table in <u>Section 12.6.3</u> ("Safety") presents the Adverse Events of Special Interest (AESI) and the groups of terms that they comprise. AESI which are not standardized MedDRA queries (SMQs) comprise a selection of PTs defined by GSK. The final list of AESIs, and the PTs that contribute to each of the AESIs, will be provided by Safety and Medical Governance (SMG), using the MedDRA version current at the time of reporting. This list will be finalized prior to unblinding the database.

Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting. Furthermore, emerging data from on-going studies may highlight additional AESI. Therefore, the list of AESI, and the terms included for each AESI, will be based on the safety review team (SRT) agreements in place at the time of reporting. The details of the planned displays are provided in <a href="Appendix 11">Appendix 11</a>: List of Data Displays.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, Lipids and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in <u>Appendix 11</u>: List of Data Displays.

A line plot of the mean change from baseline (latest pre-dose value including unscheduled visits) as well as +/- standard error over time (day) for each treatment by gender will be plotted for below mentioned sex hormones and metabolic analytes.

#### Sex / Reproductive Hormones

Testosterone, Free Testosterone, Sex hormone-binding globulin (SHBG), Follicle-stimulating hormone (FSH), Luteinizing hormone (LH) and Prostate specific antigen (PSA).

#### Metabolic Analytes

Total Cholesterol, LDL Cholesterol, HDL Cholesterol, Triglyceride, Glucose and HbA1c.

#### 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 11: List of Data Displays.

A listing of changes from baseline in hepatic, prostate (males) and cardiac structure and function assessed via MRI scan will be presented as an exploratory analysis.

Biomarkers will be summarized descriptively. The reproductive tissue biomarkers and bone markers to summarize are given below.

#### Reproductive Tissue Biomarkers

Luteinizing hormone, Follicle stimulating hormone, Total testosterone, Free testosterone (calculated) in males and female, Estradiol (females), Dihydrotestosterone, Sex hormone binding globulin and Prostate specific antigen (PSA) (males).

#### Bone Biomarkers

Procollagen type I N propeptide (s-PINP) and C-terminal telopeptide of type I collagen (s-CTX).

#### 9. PHARMACOKINETIC ANALYSES

PK concentration related summaries will be presented. No PK parameters will be derived in this RAP. The PK parameters for the Study will be derived as a part of Population Pharmacokinetic (POPPK) analyses. The POPPK RAP will include the detailed population PK analysis and resulting derived PK parameters including Cmax and AUC over dosing interval.

# 9.1. Secondary Pharmacokinetic Analyses

#### 9.1.1. Summary Measure

Pharmacokinetic concentration data will be presented in graphical and tabular form and will be summarized descriptively by gender.

#### 9.1.2. Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 9.1.3. Statistical Analyses / Methods

Details of the planned displays are provided in <u>Appendix 11</u>: List of Data Displays and will be based on GSK Data Standards and statistical principles.

#### 9.1.3.1. Statistical Methodology Specification

Plasma concentration time data will be descriptively summarized by the 3 sampling intervals (pre dose, 1-4h interval and 5-8 h intervals) by visit and also listed by treatment group for each gender.

# 10. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

A population PK analysis will be conducted on the final data. The timeline for these analyses will be independent of the analysis described in this RAP. To support this analysis a NONMEM-specific data file will be generated, the analysis approach and specifications are detailed in the POP PK Data Analysis Plan by CPMS.

To support this analysis two NONMEM-specific data files will be generated by S&P using predefined formatted datasets provided by CPMS. The first formatted dataset will focus on the PK data and all relevant covariates. The second dataset will contain the time dependent efficacy and safety endpoints.

# 11. REFERENCES

Celli BR, MacNee W, Agusti A, Anzueto A, Berg B, Buist AS, et al. Standards for the diagnosis and treatment of patients with COPD: a summary of the ATS/ERS position paper. Eur Resp J 2004 23: 932-946

IMI PROACTIVE IN COPD DAILY AND CLINICAL INSTRUMENTS D-PPAC and C-PPAC USER GIDE (14June2016)

Jones, PW and Forde Y (2016). St. Georges Respiratory Questionnaire for COPD Patients Manual, version 1.3.

Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL et al. Multi-ethnic reference values for spirometry for the 3-95 year age range: the global lung function 2012 equations. Eur Resp J. 2012; 40: 1324-1343

#### 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

#### 12.1.1. Exclusions from Per Protocol Population

The criteria for subject exclusion from the Per Protocol population are based on 'the Protocol Deviation Specification-version 2.0-31August 2018'. Refer to the latest version of the rules document prior to finalisation of the per protocol population.

The following criteria define the protocol deviations Potential protocol deviations leading to exclusion from PP population will be reviewed by the study team to confirm that they meet these criteria. This review will occur before the clinical database has been frozen for analysis. Note: None of the protocol deviations need the data unblinding to take the decision whether the subject data to be excluded from analysis or not. So, the protocol deviation meeting post unblinding won't be conducted.

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|---|---|
| 01 | Inclusion #1 – Subject not 50-75 years of age inclusive |
| 02 | Inclusion #3 – Did not have Confirmed Diagnosis of COPD |
| 03 | Inclusion #4 – SPPB: Score of "0" on any component of the SPPB or Timed Chair Stand Score is < 1 and > 3 |
| 04 | Inclusion #5 – BMI not within 18-32 kg/m2 (inclusive) |
| 05 | Inclusion #6 – not current smokers or former smokers with a cigarette smoking history of <10 pack years |
| 06 | Exclusion #1-7 – Prohibited Medical Conditions |
| 07 | Exclusion #8-10 – Prohibited Treatments |
| 08 | Exclusion #11 – Prohibited Prior/Current Clinical Study Experience |
| 09 | Exclusion #12-13 – Key laboratory tests out of range |
| 10 | Exclusion #14 – ECG values above ranges (QTc > 480, QTcB/F > 450) |
| 11 | Exclusion #15 – Positive HIV antibody test |
| 12 | Any other deviations from inclusion/exclusion criteria which could impact the efficacy assessment. |
| 13 | Experience an exacerbation, which needed treatment with steroids during the treatment phase of the study |
| 14 | Not completing the Day 80 PROactive endpoint, Week 13 (Day 90) lean mass and all of the functional assessments (leg press strength, peak performance from Incremental shuttle walking test, Constant Work Rate (CWR) duration from endurance shuttle walking test, total SPPB score and handgrip strength). |
| 15 | Permanent discontinuation of the treatment during the study treatment period (This check must will be performed by Statistics and Programming). |

# 12.2. Appendix 2: Schedule of Activities

# 12.2.1. Protocol Defined Schedule of Events

| Procedure | Screening<br>V1 | V2 | | 1 | Freatme | nt Peri | od (13 | weeks) | | Follow- | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | (up to 30<br>days before<br>Day 1) | <b>V2</b><br>Day -9 | V3<br>Baseline<br>Day 1 | V4<br>Day<br>14 | V5<br>Day<br>28 | V6<br>Day<br>56 | V7<br>Day<br>80 | V8<br>Last<br>dose<br>90 | Unscheduled<br>visit <sup>1</sup> | V9<br>(42 days<br>post last<br>dose) | |
| Visit window (days) | - 30 to -11 | -11 to<br>-7 | -2 to day<br>1 | 12 -<br>16 | 24 –<br>32 | 52-<br>60 | 76 -<br>84 | 85 –<br>91 | | 126- 140 | There should be an attempt to conduct all assessments for a visit within a single day <sup>3</sup> . |
| Informed consent | Х | | | | | | | | | | Obtained prior to performing any study-related procedures. |
| Inclusion and exclusion criteria | Х | | | | | | | | | | , , |
| Demography/ medical/medication/<br>drug/ alcohol history/ PD disease<br>staging | Х | | | | | | | | | | |
| Full physical examination | Х | | | | | | | | Х | Х | |
| Brief physical exam | | | Х | Х | Х | Х | | Х | | | |
| 12-lead ECG | Х | | Х | Х | Х | Х | | Х | Х | Х | |
| Vital signs | Х | | Χ | Χ | Χ | Χ | | Χ | Х | Х | |
| HIV, Hepatitis B and C screening | Х | | | | | | | | | | If test otherwise performed within 3 months prior to first dose of study treatment, testing at screening is not required |

| Procedure | Screening | 1/0 | Treatment Period (13 weeks) | | | | | | Follow- | Notes | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | V1<br>(up to 30<br>days before<br>Day 1) | <b>V2</b><br>Day -9 | V3<br>Baseline<br>Day 1 | V4<br>Day<br>14 | V5<br>Day<br>28 | V6<br>Day<br>56 | V7<br>Day<br>80 | V8<br>Last<br>dose<br>90 | Unscheduled<br>visit <sup>1</sup> | up <sup>2</sup><br>V9<br>(42 days<br>post last<br>dose) | |
| Hepatitis C viral RNA PCR | | | | | | | | | X | | If evidence of Hepatitis C antibodies at screening visit, then Hepatitis C viral RNA PCR required to exclude active infection. This sample is not needed if Hepatitis C screening is negative. |
| Haematology (Full blood count)/<br>Clinical Chemistry (Creatinine, urea<br>and electrolytes, liver function tests,<br>glucose) | Х | | Х | Х | Х | Х | | Х | Х | Х | Participants should fast overnight for at least 8 hours prior to collection of these samples. |
| HbA1c | Χ | | | | | | | Х | | | |
| hsCRP, Fibrinogen | | | Х | | | | | Χ | | Х | |
| 25-OH Vitamin D Total, 25-OH<br>Vitamin D2, 25-OH Vitamin D3 | X | | | | | | | Х | | Х | |
| Lipid panel | X | | Χ | Χ | Χ | Χ | | Х | | Χ | |
| Genetic sample | | | Х | | | | | | | | Obtain after participant is randomized. <b>Informed consent to obtain the genetics sample</b> must be obtained before collecting a sample. |
| Pharmacokinetic sampling | | | | X <sup>4</sup> | X <sup>4,5</sup> | X6 | | X <sup>4</sup> | X | | Times of dose administration for the two doses immediately preceding a PK sample should be accurately recorded. |
| Reproductive Tissue Biomarkers | | | Х | | Χ | Χ | | Х | | Х | |
| PSA | Х | | Х | | Χ | Χ | | Х | | Х | For male participants only |
| Bone Biomarkers | | | Χ | | | Χ | | Χ | | Х | |
| V1 (up to 30 days before Day 1) Exploratory Biomarkers Urinalysis X DXA Spirometry X Sniff Nasal Inspiratory Pressure X Leg strength X Handgrip strength X Short Physical Performance Battery X Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical Activity Monitor | | <b>V2</b> Day -9 | V3<br>Baseline<br>Day 1 | V4<br>Day<br>14 | V5<br>Day | V6 | \/7 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Urinalysis X DXA Spirometry X Sniff Nasal Inspiratory Pressure X Leg strength X Handgrip strength X Short Physical Performance Battery X Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical | | | | | 28 | Day<br>56 | V7<br>Day<br>80 | V8<br>Last<br>dose<br>90 | Unscheduled<br>visit <sup>1</sup> | up <sup>2</sup><br>V9<br>(42 days<br>post last<br>dose) | |
| Spirometry Sniff Nasal Inspiratory Pressure Leg strength X Handgrip strength Short Physical Performance Battery Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | Χ | Χ | Χ | | Χ | | Χ | |
| Spirometry Sniff Nasal Inspiratory Pressure Leg strength X Handgrip strength X Short Physical Performance Battery Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | | | | | Χ | Χ | X | |
| Sniff Nasal Inspiratory Pressure X Leg strength X Handgrip strength X Short Physical Performance Battery X Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Х | | Χ | Χ | | Χ | Χ | Χ | |
| Leg strength X Handgrip strength X Short Physical Performance Battery X Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Х | | | Х | | Х | | | Follow ATS/ ERS guidelines [Celli, 2004] and Quanjer reference equation [Quanjer, 2012]. |
| Handgrip strength X Short Physical Performance Battery X Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | | | Χ | | Χ | | | |
| Short Physical Performance Battery Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | | Χ | Χ | | Χ | | Χ | |
| Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | | | | | Χ | | | |
| Incremental Shuttle Walk Test Endurance Shuttle Walk Test COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | | Χ | Χ | | Χ | | Х | |
| COPD Assessment Test St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | Х | Х | Х | | | | | Χ | | | Practice incremental shuttle walk test conducted at day -9 |
| St George Respiratory Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | | | | | Χ | | | |
| Questionnaire COPD (SGRQ-c) Patient Global Rating of Severity Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | | | Χ | | Χ | | | |
| Patient Global Impression of Change Daily PROactive Physical Activity in COPD instrument and Physical X | | | Х | | | | | Χ | | | |
| Daily PROactive Physical Activity in COPD instrument and Physical X | | | Χ | | | | | Χ | | | |
| COPD instrument and Physical X | | | | Х | Χ | Χ | | Χ | | Χ | |
| Productly Mornton | X <sup>7</sup> | X <sup>7</sup> | | | | Χ | <b>X</b> <sup>7</sup> | | | | Physical activity monitor dispensed at screening, day -9, day 56 and day 80 visits. Activity monitor should be worn for 7 days at each timepoint and returned at the next visit. |
| Monitored home exercise program Patient exit interview | Х | х | Х | <b>←==</b> | ===== | ==== | ==-> | Х | | X | Participants will receive training for<br>the exercise program at Day -9,<br>and will formally begin exercises<br>on day 1 |

| Procedure | Screening<br>V1 | V2 | | 1 | reatme | nt Peri | od (13 | weeks) | | Follow- | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | (up to 30<br>days before<br>Day 1) | Day -9 | V3<br>Baseline<br>Day 1 | V4<br>Day<br>14 | V5<br>Day<br>28 | V6<br>Day<br>56 | V7<br>Day<br>80 | V8<br>Last<br>dose<br>90 | Unscheduled<br>visit <sup>1</sup> | V9<br>(42 days<br>post last<br>dose) | |
| Randomization | | | Х | | | | | | | | All Baseline assessments must be obtained prior to randomization. |
| Study treatment provided to participant | | | Х | | Х | Х | | | | | The subject should take their first dose of study treatment in the clinic after randomization. |
| Study treatment | | | Х | <b>←==</b> | ===== | ===== | ==→ | Х | | | Participants should dose study treatment in the clinic at each clinic visit during the treatment period. |
| Study treatment accountability by study site | | | Х | Х | Х | Х | | Х | | | The required counting of pills by site staff to check compliance is not considered redispensing the study medication. |
| AE review | | | Χ | + | <del>-===</del> | | | ===== | =====> | Х | |
| SAE review | | | Χ | • | <del>(</del> ==== | | | ===== | =====→ | Χ | |
| Concomitant medication review | | | Χ | • | <del>(</del> ==== | ===== | ===== | ===== | =====→ | Х | |
| Optional sub-study measures | | | | | | | | | | | |
| Cardiac and liver MRI (additionally prostate MRI in males) | | | X8 | | | | | X8 | | | MRI is an optional assessment undertaken at participating centres only. |

ECG= Electrocardiogram; HIV= Human Immunodeficiency Virus; PK= Pharmacokinetic; PSA= Prostate Specific Antigen; DXA= Dual-energy X-ray Absorptiometry; AE= Adverse Event; SAE= Serious Adverse Event.

1. An unscheduled clinic visit may occur at any time if the investigator believes an unscheduled visit is clinically warranted. Individual listed assessments are optional and are performed as needed to follow unresolved findings of clinical concern. Note: The "Unscheduled visit" case report form (CRF) form should be completed as soon as possible following the Unscheduled visit.

- 2. As stated in Section 8.2, if a participant decides to withdraw or is withdrawn by the responsible physician, the reasons for withdrawal and the results of any relevant tests will be recorded in the CRF and the planned safety follow-up procedures will be performed, where possible. These include physical examination, 12-lead ECG, vitals, blood tests, urinalysis and concomitant medication review as listed for the follow-up visit (V9).
- 3. Attempt to conduct all visits within a single day however the baseline (day 1) and last dose (day 90) visits may require subjects to visit the study centre on more than one day in order to complete MRI and DXA scans, and possibly other assessments. These scans, and any other assessments, should be conducted within the specified visit window, and prior to randomization at the baseline visit. Further details on the suggested order of assessments will be given in the SRM.
- 4. Take PK sample prior to dosing in the clinic
- 5. Take PK sample 1-4 hours post-dose (sites should try and ensure that a range of times are sampled within this time window for different participants, i.e. all PK samples should not be taken at 1 hour post dose or 2 hours post dose).
- 6. Take PK sample 5-8 hours post-dose (as above, sites should try and ensure that a range of times are sampled within this time window for different participants).
- 7. At V3 Baseline Day 1 and V8 Last dose 90, the patients will return the Daily PROactive Physical Activity in COPD Instrument and the Physical Activity Monitor to the site. Patients will not be dispensed the Daily PROactive Physical Activity in COPD Instrument and the Physical Activity Monitor at the end of these visits.
- 8. All MRI Scans (Cardiac MRI, Liver MRI and, if applicable, Prostate MRI) should preferably be scheduled on the same day. Acquisition of the Cardiac MRI should be prioritized above the other two scans if it becomes unfeasible to perform all the MRI scan.

The following points must be noted:

- If assessments are scheduled for the same nominal time, THEN the assessments should occur in the following order:
  - i. vital signs
  - ii. 12-lead ECG
  - iii. blood draws.

Note: The timing of the assessments should allow the blood draw to occur at the time specified in the SoA.

## 12.3. Appendix 3: Assessment Windows

## 12.3.1. Definitions of Assessment Windows for Analyses

| Analysis | Parameter | Protocol Wi | indow | Target | Analysis | Window | Analysis |
|---|---|---|---|---|---|---|---|
| Set /<br>Domain | (if applicable) | Beginning<br>Timepoint | Ending<br>Timepoint | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| All | All | Day -30 | Day -11 | Day -<br>30 to -<br>11 | Day -60 | Day -12 | Screening/Visit<br>1 |
| All | All | Day -11 | Day -7 | Day -9 | Day -11 | Day -5 | Visit 2 |
| All | All | Day -2 | Day 1 | Day 1 | Day -4 | Day 1 | Visit 3, Day 1 |
| All | All | Day 12 | Day 16 | Day 14 | Day 10 | Day 18 | Visit 4, Day 14 |
| All | All | Day 24 | Day 32 | Day 28 | Day 22 | Day 34 | Visit 5, Day 28 |
| All | All | Day 52 | Day 60 | Day 56 | Day 50 | Day 62 | Visit 6, Day 56 |
| All | All | Day 76 | Day 84 | Day 80 | Day 76 | Day 84 | Visit 7, Day 80 |
| All | All | Day 85 | Day 91 | Day 90 | Day 85 | Day 97 | Visit 8, Day 90 |
| All | All | Day 126 | Day 140 | Day<br>132 | Day 126 | Day 140 | Follow-Up, Day<br>132 |

- For scheduled visits the analysis visit would equal the nominal visit irrespective of the assessment date and irrespective of whether that date falls in the visit window.
- Only unscheduled visits are slotted according to the table above and this slotting algorithm will be applicable for both efficacy and safety domains.
- After slotting of Un-scheduled visits, if there are multiple assessments at a planned timepoint, then the value closest to the target day for that window will be considered. If the multiple assessments are equidistant from the target day, then mean of the assessments will be considered.
- For any time post baseline and baseline (if the definition of baseline is the latest pre-dose visit) all assessments are used irrespective of whether they fall into visit windows or not.

## 12.4. Appendix 4: Study Phases

## 12.4.1. Study Phases

Only Concomitant Medication will be reported by treatment phases and all other displays will be irrespective of the phases.

## 12.4.2. Study Phases for Concomitant Medication

| Definition | Treatme | Treatment Phase |
|---|---|---|
| Definition | Pre-Treatment | On-Treatment* |
| Subject did not take study treatment (e.g., screening failures) AND concomitant medication stop date >= date of Screening | Y | |
| Concomitant medication start date < treatment start date AND (date of Screening <= concomitant medication stop date <treatment date)<="" start="" td=""><td>Y</td><td></td></treatment> | Y | |
| Concomitant medication start date < (treatment start date or screening Date) and the variable that defines the status of Concomitant medication end with respect to reference time -period is ("BEFORE") | Y | |
| Concomitant medication start date < treatment start date AND the variable that defines the status of Concomitant medication end with respect to reference time -period is ("AFTER", "DURING", "DURING/AFTER", "ONGOING") | Y | Υ |
| Concomitant medication start date < treatment start date AND (treatment start date < concomitant medication stop date <= treatment stop date) | Y | Υ |
| (Concomitant medication start date < treatment start date) AND (concomitant medication stop date > treatment stop date) | Y | Υ |
| Treatment start date <= concomitant medication start date | | Υ |

<sup>\*</sup>On-Treatment phase includes both On-Treatment and Post-Treatment concomitant medications.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

## 12.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently supply | The currently supported versions of SAS software (Version 9.2 or higher). |
| Reporting Area | |
| HARP Server | : us1salx00259 |
| HARP Compound : \ARPROD\GSK2881078\mid200182\ | |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & AdaM IG Version 1.0. | |

For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be

# implemented as SDTM. Generation of RTF Files

RTF files will be generated for each reporting effort.

## 12.5.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF except for the parameters specified below.

| Domain | DP for Mean |
|---|---|
| Leg Press (Last Successful Lift 1-Rep Max (kg)) | 1 DP |
| Appendicular Lean Mass (kg) & Total Lean Mass (kg) | 3 DP |
| PRO parameters & SGRQ parameters | 2 DP |
| Total Score for SPPB | 1 DP |
| CAT | 1 DP |
| Time for the Fastest Walk (sec) & Time Repeated Chair Stand Test (sec) | 3 DP |

| Incremental Shuttle Walking test - Maximum Distance Walked (m) | 1 DP |
|----------------------------------------------------------------|------|
| CWR - Exercise Duration (sec) | 1 DP |

 The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using the assessment windows defined in <u>Section 12.3</u>. After slotting of Un-scheduled visits, if there are multiple assessments at a planned time-point, then the value closest to the target day for that window will be used. If its equidistant from the target day, then mean of the assessments will be used in summary and figures. Listing will show both the planned and un-scheduled assessments.
- Data summaries will only report visits that are planned assessment time points for each parameter (according to the T&E table) which can include the unscheduled visits if slotted.
- All unscheduled visits will be included in listings.
- Unscheduled visits can be included in the derivation of any time post baseline visits and baseline if the definition of baseline is the latest pre-dose visit (See Section 5.2).

| Descriptive Summary Statistics |
|------------------------------------------------------------|
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data N, n, frequency, % |
| Graphical Displays |
| Refer to IDSL Statistical Principals 7.01 to 7.13. |

## 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements (not in case of visit slotting) will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per <u>Section 12.3.1</u>) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

Note that Treatment Start Date is considered as Study Day 1.

#### Post-baseline

Post-baseline refers to the combined time periods of On-treatment and Post-treatment.

## **Change from Baseline**

= Post-baseline -Baseline

#### Ratio to Baseline

= exp (log (Post-baseline) -log (Baseline))

#### **Percent Change from Baseline**

= 100\*(Post-baseline – Baseline)/Baseline

#### Treatment compliance

= 100 \* (Total Amount Taken/ (Treatment duration in days\* 2))

Total Amount Taken = Total tablets dispensed – Total tablets returned – Total tablets lost.

## 12.6.2. Efficacy

## **Secondary Efficacy endpoints**

## Peak performance from incremental shuttle walking test

'Maximum distance walked' collected from incremental shuttle walk test in CRF

#### Constant Work Rate (CWR) duration from endurance shuttle walking test

'Exercise duration time (seconds)' collected from endurance shuttle walk test in CRF

## St George Respiratory Questionnaire (SGRQ) total score and domains

 The total score and three component scores (Symptoms, Activity and Impacts) will be derived from St George Respiratory Questionnaire- COPD (SGRQ- c) raw scores based upon the score manual (ST

#### **Secondary Efficacy endpoints**

GEORGE'S RESPIRATORY QUESTIONNAIRE FOR COPD PATIENTS (SGRQ-C) Version No.1.3 March 2016)

• First, sum the weights for all items with a positive response:

Symptoms component consists of all the questions (question 1 -7) in Part 1. The weights for Questions 1-7 are summed. A single response is required to each item. If multiple responses are given to an item, the weights for the multiple positive responses should be averaged then added to the sum.

Activity component is calculated from the summed weights for the positive responses to items questions 9 and 12 in Part 2 of the questionnaire.

Impacts component is calculated from questions 8, 10, 11, 13, 14 in Part 2 of the questionnaire. The weights for all positive responses to items in Questions 10, 11, 13 are summed together with the responses to the single item that should have been checked (ticked) in Questions 8 and 14. In the case of multiple responses to either of these items, the average weight for the item should be calculated.

Total score is calculated by summing the weight to all the positive responses in each component.

• Then, calculate the score:

The score for each component is calculated separately by dividing the summed weights by the maximum possible weight for that component and expressing the results as a percentage: Sum of maximum possible weights for each component and Total:

Symptoms: 566.2 Impact: 1652.8 Activity: 982.9 Total: 3201.9

Last, converting SGRQ-c scores to be comparable to SGRQ:

The adjustment is:

Symptoms: SGRQ score = (SGRQ-C x 0.99) + 0.94 units Activity: SGRQ score = (SGRQ-C x 0.87) +7.01 units Impacts: SGRQ score = (SGRQ-C x 0.88) +2.18 units Total: SGRQ score = (SGRQ-C x 0.90) + 3.10 units

#### Handling of missing items

A Total score can be calculated in the presence of missing data, but only if the domains meet their 'missing items' rules (see below). If one domain exceeds its permitted number of missed items, then a total score cannot be calculated.

Symptoms: The Symptoms component will tolerate a maximum of 1 missed item. The weight for the missed item is subtracted from the total possible weight for the Symptoms component (566.2) and from the Total weight (3201.9) and then calculate the score.

Activity: The Activity component will tolerate a maximum of 3 missed items. The weight for the missed item (s) is subtracted from the total possible weight for the Activity component (982.9) and from the Total weight (3201.9) and then calculate the score.

Impacts: The Impacts component will tolerate a maximum of 5 missed items. The weight for the missed item (s) is subtracted from the total possible weight for the Impacts component (1652.8) and from the Total weight (3201.9) and then calculate the score.

• Responder is defined as 'Yes' when the total score at a post-baseline visit decreases by 4 or more from baseline total score, otherwise, non-responder.

## **Secondary Efficacy endpoints**

# Total Short Physical Performance Battery (SPPB) score and times for chair rise and 4 m gait speed

- Total SPPB score, 'Time for five stands done successfully' collected for chair and 'time for fastest walk for 4 m gait test' collected from CRF will be used, respectively
- SPPB at baseline will be categorized as below:

SPPB 10-12 points fit patient, normal

SPPB 8-9 points pre-frail patient

SPPB ≤ 7 points frail patient

### **COPD Assessment Test (CAT)**

- Total score of 8 questions will be used
- Responder is defined as 'Yes' when the total score at a post-baseline visit decreases by 2 or more from baseline total score, otherwise, non-responder.
- If one or more of the 8 questions are missing the total score and the responder will be missing.

## PROactive endpoints (individual components (Difficulty and Amount) and total score)

- The PROactive instrument (IMI PROACTIVE IN COPD DAILY AND CLINICAL INSTRUMENTS D-PPAC and C-PPAC 2016 (Use D-PPAC for the calculation of scores)) combines a PRO questionnaire and an activity monitor to measure physical activity in COPD patients. It is 9-item daily assessments covering 2 different domains (amount and difficulty) designed for electronic administration. The 'amount' domain is covered by 2 items (questions amount of walking outside and chores outside) and by 2 activity monitor outputs (vector magnitude units per minute (VMU/min) and steps/day). The 'difficulty' domain is covered by 5 items (questions).
- The scores for activity monitor outputs, step counts and VMU's is assigned based on the 5 level categories they are falling in (see the table below).

Scores

VMU/min

Steps/day

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

Calculation of daily score for each domain (amount, difficulty) and total score:
 First, domains are scored by simple adding items, which, the values are 0-17 for 'amount' and 0-20 for 'difficulty'. The raw scores are then scaled to a score ranging from 0 to 100, based on Table 1 in the guidance (see Reference)

The 'total score' is obtained calculating the average between two domains. This score has the same scale of two individual domains, from 0 to 100.

PROactive scores for a day cannot be calculated if the subjects missed any of the 9 items in any day.

## Secondary Efficacy endpoints

- Calculation of the weekly score for each domain (amount, difficulty) and total score:
   The average of the daily scores during a 7-day period will be the weekly score separately for each domain (amount, difficulty) and total score.
- Score eligibility:

Adequate physical activity data are considered for days where more than eight hours of wearing time is available. The activity monitor measurement days used should be concurrent with the questionnaire.

At least four days with  $\geq 8$  hours of wearing time of activity monitor data are required for the measurements to be valid for a weekly average. These four days should be in the same week (7 days from the first day of assessments), do not need to be consecutive, and could cover weekdays or weekend days without distinction.

#### **Physical Activity Measures**

- At least four days with ≥ 8 hours of wearing time of activity monitor data are required for the
  measurements to be valid for a weekly average. These four days should be in the same week (7 days
  from the first day of assessments), do not need to be consecutive, and could cover weekdays or
  weekend days without distinction. Then calculate the average by dividing total with number of days.
- The physical activity measures weekly average steps, weekly average vector magnitude unit/wear time and weekly average moderate/vigorous activity duration have the same derivation.
- The number of subjects included: The count of subject in each visit who has wear time more than 8 hours for at least 4 days in a week.
- Average number of days included per subject: This the average number of days with wear duration more than 8 hours for at least 4 days in each visit.
- Average number of minutes included per subject: This the average wear duration in minutes for those subjects with more than 8 hours of wear duration for at least 4 days in a week for each visit.

## 12.6.3. Safety

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

Duration of Exposure in Days = Treatment Stop Date – (Treatment Start Date) + 1
The number of days exposure therefore does not take into account dose interruptions.

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- Actual amount taken (number of tablets) = Total tablets dispensed Total tablets returned Total tablets lost.
- Females will take 1 mg everyday (2\*0.5mg tables) and males will take 2 mg (2\*1mg). So, the actual dose (mg) taken will be the same as actual amount taken for males and for females it will be actual amount taken divided by 2.
- The cumulative actual dose (mg) will be the sum of the actual doses taken.

| Adverse Events | |
|---|---|
| Onset Time Since | If Treatment Start Datetime ≤ AE Onset Datetime , then AE Onset Datetime - |
| 1st Dose (Days) | Treatment Start Datetime +1 |
| | If time part is missing in any of the Datetime, then use the Treatment Start date and AE |

| Extent of Exposur | Extent of Exposure |
|---|---|
| | Onset date in calculation and missing otherwise. |
| Duration (Days) | AE Resolution Datetime – AE Onset Datetime + 1 |
| | If time part is missing in any of the Datetime, then use the AE Resolution date and AE |
| | Onset date in calculation and missing otherwise. |
| Drug-related | If the question 'is there a reasonable possibility that AE may have been caused by the |
| | Study Treatment' is marked 'YES' on CRF or is missing. |

#### MRI

- Body Surface Area (BSA) (m<sup>2</sup>) =0.007184 \* Weight (kg)<sup>0.425</sup> \* Height (cm)<sup>0.725</sup>
- Left Ventricular End Systolic Volume Index (LVESVi)=
   LVESV

Body Surface Area

Left Ventricular End Diastolic Volume Index (LVEDVi)= LVEDV

Body Surface Area

## **Adverse Events**

## Adverse Events of Special Interest (AESI))

The following table presents the AESI. AESI which are not SMQs are made up of a selection of preferred terms (PTs) defined by GSK. The complete list of AESI, including the PTs which contribute to each of the AESI will be provided by Safety and Medical Governance using the MedDRA version current at the time of reporting.

| AESI | Group of terms (MedDRA | SMQ, HLT or individual PTs) |
|---|---|---|
| Drug related hepatic disorders | Drug related hepatic disorders – comprehensive search (SMQ) | |
| Reproductive organ | Prostatic neoplasms and hypertrophy HLT plus selected preferred terms: | |
| effects, male | Prostatic specific antigen abnormal | |
| | Prostatic specific antigen increased | |
| Reproductive organ effects, female | Female gonadal function disorders HLT (includes PT of Hirsutism and Virilism) | |
| Virilism in females | Hirsutism PT, Virilism PT, Acnes HLT, Dysphonia PT | |
| Dyslipidaemia | Dyslipidaemia SMQ | |
| Bone effects | Osteoporosis/osteopenia (SMQ), | |
| | Plus, selected Fracture PTs (57 terms) | |
| | MedDRA PT | PT Code |
| | Ankle fracture | 10002544 |
| | Bone decalcification | 10070817 |
| | Bone disorder | 10005956 |
| | Bone fragmentation | 10064211 |
| | Clavicle fracture | 10009245 |
| | Comminuted fracture | 10052614 |
| | Complicated fracture | 10010149 |
| | Compression fracture | 10010214 |

| Expiphyseal fracture | | |
|---|---|---|
| Fibula fracture | Epiphyseal fracture | 10053962 |
| Fracture delayed union | Facial bones fracture | 10016042 |
| Fracture delayed union | Fibula fracture | 10016667 |
| Fracture displacement | Foot fracture | 10016970 |
| Fracture reduction | Fracture delayed union | 10017081 |
| Fracture reduction | Fracture displacement | 10053206 |
| Fractured skull depressed | | 10057609 |
| Fractured skull depressed | Fractured coccvx | 10049164 |
| Greenstick fracture | 1 | |
| Hand fracture | · | |
| Humerus fracture | | |
| Impacted fracture | | |
| Internal fixation of spine | | |
| Jaw fracture | | |
| Lower limb fracture | · | |
| Open fracture 10030527 Osteocalcin decreased 10050940 Osteonecrosis 10031264 Osteonecrosis of jaw 10064658 Patella fracture 10034122 Scapula fracture 10039579 Skeletal injury 10061363 Skull fracture 10061365 Skull fractured base 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10074807 Fracture malunion 10017088 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening | | |
| Osteocalcin decreased 10050940 Osteonecrosis 10031264 Osteonecrosis of jaw 10064658 Patella fracture 10034122 Scapula fracture 10039579 Skeletal injury 10061363 Skull fracture 10061365 Skull fractured base 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 1007395 Avulsion fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Osteonecrosis 10031264 Osteonecrosis of jaw 10064658 Patella fracture 10034122 Scapula fracture 10039579 Skeletal injury 10061363 Skull fracture 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 1007395 Avulsion fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077956 Bone metabolism biochemical marker increased 10078949 | | |
| Osteonecrosis of jaw 10064658 Patella fracture 10034122 Scapula fracture 10039579 Skeletal injury 10061363 Skull fracture 10061365 Skull fractured base 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10073551 Osteochondral fracture 10073853 Periprosthetic fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Patella fracture 10034122 Scapula fracture 10039579 Skeletal injury 10061363 Skull fracture 10040960 Stull fractured base 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10073853 Periprosthetic fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Scapula fracture 10039579 Skeletal injury 10061363 Skull fracture 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 1007351 Osteochondral fracture 100793853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077756 Bone metabolism biochemical marker increased 10078949 | <del> </del> | |
| Skeletal injury 10061363 Skull fracture 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10066094 Traumatic fracture 10045375 Ulna fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Skull fracture 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 1007352 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Skull fractured base 10040960 Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077956 Bone metabolism biochemical marker increased 10078949 | | |
| Sternal fracture 10042015 Stress fracture 10042212 Tibia fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10073162 Limb fracture 10073162 Limb fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 100778949 increased 10078949 | | |
| Stress fracture 10042212 Tibia fracture 10043827 Torus fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Tibia fracture 10043827 Torus fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Torus fracture 10066094 Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Traumatic fracture 10049514 Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Ulna fracture 10045375 Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077756 Bone metabolism biochemical marker increased | | |
| Upper limb fracture 10061394 Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Vertebral wedging 10065317 Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Atypical fracture 10072395 Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Avulsion fracture 10066184 Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10069135 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Chance fracture 10073162 Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Limb fracture 10074551 Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Osteochondral fracture 10073853 Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | |
| Periprosthetic fracture 10069135 Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | | 10074551 |
| Spinal fusion fracture 10074807 Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | Osteochondral fracture | 10073853 |
| Fracture malunion 10017085 Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | Periprosthetic fracture | 10069135 |
| Fracture nonunion 10017088 Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | Spinal fusion fracture | 10074807 |
| Craniofacial fracture 10077603 Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | Fracture malunion | 10017085 |
| Spinal flattening 10077756 Bone metabolism biochemical marker increased 10078949 | Fracture nonunion | 10017088 |
| Bone metabolism biochemical marker 10078949 increased | Craniofacial fracture | 10077603 |
| Bone metabolism biochemical marker 10078949 increased | Spinal flattening | 10077756 |
| | | 10078949 |
| Subchondral insufficiency fracture 10079864 | increased | |
| | Subchondral insufficiency fracture | 10079864 |

| | Maisonneuve fracture | 10081343 |
|---|---|---|
| | Degenerative bone disease | 10081730 |
| | Internal fixation of fracture | 10022576 |
| Cardiovascular effects | See the table below. | |
| Hypersensitivity | Hypersensitivity (SMQ) narrow, Angioedema (SMQ) narrow, Anaphylactic reaction (SMQ) narrow | |
| Hostility/aggression | Hostility/aggression (SMQ) | |
| Sexual desire disorders | Sexual desire disorders HLT | |
| Embolic and thrombotic events | Embolic and thrombotic events (SMQ) | |

## **Cardiovascular effects AESI**

| AESI | AESI Subgroup | Sub-SMQ | Scope |
|---|---|---|---|
| Cardiovascular Cardiac arrhythmia effects | | Arrhythmia related investigations, signs and symptoms (SMQ) | Broad |
| | | Bradyarrhythmia terms, nonspecific (SMQ) | Broad |
| | | Conduction defects (SMQ) | Broad |
| | | Disorders of sinus node function (SMQ) | Broad |
| | | Cardiac arrhythmia terms, nonspecific (SMQ) | Broad |
| | | Supraventricular tachyarrhythmias (SMQ) | Broad |
| | | Tachyarrhythmia terms, nonspecific (SMQ) | Broad |
| | | Ventricular tachyarrhythmias (SMQ) | Broad |
| | Cardiac failure (SMQ) | | Broad |
| | Ischaemic heart disease (SMQ) | | Broad |
| | Hypertension (SMQ) | | Broad |
| Central nervous system haemorrhage and cerebrovascular conditions (SMQ) | | | Broad |
| | Cardiomyopathy (SMQ) | | Narrow |

## **ECG Parameters**

## General

 The summary should be based on average value of triplicate ECG readings obtained over a brief recording period (missing readings will not be counted).

## **Eligibility Criteria**

• The QT values at screening will be using for the eligibility checking of subjects.

#### **ECG Parameters**

## **Stopping Criteria**

A subject who meet either of the bulleted criteria below will be withdrawn from the study:

- QT interval corrected for heart rate by Bazett's formula (QTcB) or QT interval corrected for heart rate by Fridericia's formula (QTcF) >450 msec
- QT interval corrected for heart rate (QTc) >480 msec in participants with Bundle Branch Block based on a single ECG.

## **Laboratory Parameters**

#### General

- All clinical laboratory tests will be based on central laboratory assessments only. If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digits = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

## **Laboratory Toxicity Grade**

- Toxicities will be based on FDA guidance 'Common Terminology Criteria for adverse events v4.03 (CTCAE) defined by NCI-CTEP (National Cancer Institute – Cancer Therapy Evaluation Program).
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the normal range.

| Parameter | Below Normal Range | Above Normal Range |
|----------------|--------------------|--------------------|
| Fasted glucose | Hypoglycaemia | Hyperglycaemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |
| Calcium | Hypocalcemia | Hypercalcemia |

## **Hepatitis Status**

- Hepatitis B and C will be determined using antibody (IgM or IgG) at the screening or within 3 months
  prior to first dose of study treatment. If there is evidence of Hepatitis C antibodies at the screening visit,
  then Hepatitis C viral RNA PCR is required to exclude active infection. This sample is not needed if
  Hepatitis C screening is negative
- Antibody (IgM or IgG) status with 'BORDERLINE' or 'REACTIVE' will be considered Positive
- A subject will be considered positive for hepatitis B virus (HBV) if they have a positive surface antigen (HBsAg) during screening. Subjects positive for HBV are not allowed to enter the study

### **COPD Exacerbation Event Count**

- The total number of exacerbation events is determined by summing the number of times there is a non-missing "Date of Onset" on the exacerbation CRF page" for a subject
- The number of exacerbating patients refers to the count of the unique patient in the COPD
   Exacerbation CRF data. In other words, it is the total number of patients who experience one or more exacerbations defied in the first bullet.

## 12.7. Appendix 7: Reporting Standards for Missing Data

## 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as subjects who completed all visits of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> <li>Withdrawal visits will be assigned to a planned visit or an unscheduled visit and will be slotted as per Appendix 3: Assessment Windows.</li> </ul> |

## 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in subject listing displays.</li> </ul> |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 12.8. Appendix 8: Values of Potential Clinical Importance

## 12.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (<<br>x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| ricinatociit | 1 | $\Delta$ from BL (Female & Male) | 0.075 | |
| | | Male | | 180 |
| Haemoglobin | g/L | Female | | 180 |
| Tidemoglobiii | | $\Delta$ from BL (Female & Male) | 25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| White Blood Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | µmol/L | $\Delta$ from BL | | 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 (Bicarbonate) | mmol/L | | 18 | 32 |

| Liver Function | | | |
|----------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | >=3xULN |
| AST/SGOT | U/L | High | >=2xULN |
| Alkaline phosphatase | U/L | High | >=2xULN |
| T Bilirubin | µmol/L | High | >=1.5ULN |
| | µmol/L | | >=1.5ULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | >=3xULN ALT |

## 12.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | • | | |
| Absolute QTc Interval | msec | N/A | > 500 |
| Uncorrected QT | msec | N/A | > 600 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | N/A | > 60 |

# 12.8.3. Vital Signs

| Vital Sign Parameter | Units | Units Clinical Concern Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | >100 |
| Pulse Rate | Beats/min | <40 | >110 |
| Respiratory Rate | breaths/min | N/A | >20 |
| Temperature (skin) | °C | N/A | >38 |

# 12.9. Appendix 9: Model Checking and Diagnostics for Statistical Analyses

# Analysis Mixed Model Repeated Measure (MMRM)

Distributional assumptions underlying the model used for analysis will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
values (i.e. checking the normality assumption and constant variance assumption of the model
respectively) to gain confidence that the model assumptions are reasonable.

## Analysis Bayesian Analysis

- Non-informative prior should be plotted to make sure it is truly non-informative.
- Adequate values for the number of MCMC samples / thinning / number of burn-in samples should be chosen to ensure that the ratio Monte Carlo Standard Errors (MCSE) and standard deviation of the posterior distribution for all the parameters in the model as small as possible, typically close to 0.01.
- In addition, if possible, the number of tuning units and maximum number of tuning iterations
  may be increased to find a better proposal distribution for the model parameters, which in turn
  may reduce the MCSE/SD ratio.
- The Geweke diagnostic test checks whether the mean estimates have converged by comparing means from the early and latter part of the Markov chain using a z score t-test.
   Large absolute values of the z-score statistic indicate rejection of the null hypothesis of no difference between the mean estimates obtained from the early and latter parts of the chain.
- The convergence diagnostics for all parameters in the Bayesian analysis will be visually checked by the trace plots.
- If the trace plots show apparent trend or the autocorrelation plots show significant positive or negative autocorrelation, number of iterations will be increased or reparameterization might be explored.

## Analysis of covariance (ANCOVA)

Distributional assumptions underlying the model used for analysis will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
values (i.e. checking the normality assumption and constant variance assumption of the model
respectively) to gain confidence that the model assumptions are reasonable.

## 12.10. Appendix 10: Abbreviations & Trade Marks

## 12.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| 1-RM | 1 repetition maximum |
| AP | Analysis Population |
| A&R | Analysis and Reporting |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | |
| BDRM | Akaike's Information Criteria |
| | Blinded data review meeting |
| BP | Blood Pressure |
| BS | Biostatistics |
| CAT | COPD Assessment Test |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| COPD | Chronic Obstructive Pulmonary Disease |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CRF | Case report form |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV | Cardiovascular |
| CVA | Cerebrovascular event stroke |
| CWR | Constant Work Rate |
| DAP | Data Analysis Plan |
| DBF | Database Freeze |
| DBR | Database Release |
| DM | Data management |
| DOB | Date of Birth |
| DP | Decimal Places |
| DVT | Deep vein thrombosis |
| DXA | Dual-energy X-ray Absorptiometry |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FSH | Follicle-stimulating hormone |
| GSK | GlaxoSmithKline |
| HR | Heart rate |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| IP | Investigational Product |
| LH | Luteinizing hormone |
| LVEF | Left ventricular ejection fraction |
| MMRM | Mixed Model Repeated Measures |
| MRI | Magnetic Resonance Imaging |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PE | Pulmonary embolism |
| PGIC | Patient Global Impression of Change |
| PGRS | Patient Global Rating of Severity |
| PSA | Prostate specific antigen |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAMOS | Randomization & Medication Ordering System |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SARM | Selective Androgen Receptor Modulator |
| SD | Standard deviation |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SE | Standard error |
| SGRQ | St George Respiratory Questionnaire |
| SGRQ-c | St George Respiratory Questionnaire-COPD |
| SMG | Safety and Medical Governance |
| SnIP | Sniff Nasal Inspiratory Pressure |
| SOP | Standard Operation Procedure |
| SPPB | Short Physical Performance Battery |
| SRT | Safety Review Team |
| SHBG | Sex hormone-binding globulin |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TIA | Transient ischemic attack |
| FEV1 | Forced Expiratory Volume in 1 second |
| SnIP | Sniff Nasal Inspiratory Pressure |

## 12.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | ( | Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|---|---|
| None | No | lone |

## 12.11. Appendix 11: List of Data Displays

## 12.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.13 | |
| Efficacy | 2.1 to 2.47 | 2.1 to 2.9 |
| Safety | 3.1 to 3.36 | 3.1 to 3.4 |
| PK | 4.1 | |
| Section | Listin | gs |
| ICH Listings | 1 to 34 | |
| Other Listings | 35 to | 89 |

## 12.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in <u>Appendix 12</u>: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 12.11.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 12.11.4. Study Population Tables

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | All<br>Participants | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | All<br>Participants | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| 1.4. | Enrolled | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Protoc | ol Deviation | | | | |
| 1.5. | All<br>Participants | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Popula | tion Analysed | | | | |
| 1.6. | Screened | SP1 | Summary of Study Populations | IDSL | Headline<br>Results & SAC |
| 1.7. | All<br>Participants | SP2 | Summary of Exclusions from the Per Protocol Population | IDSL | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.8. | All<br>Participants | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT Footnote: Age is imputed when full date of birth is not provided. | Headline<br>Results & SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.9. | Enrolled | DM11 | Summary of Age Ranges | EudraCT Footnote: Age is imputed when full date of birth is not provided. | SAC |
| 1.10. | All<br>Participants | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |
| Prior an | d Concomitan | t Medications | | | |
| 1.11. | All<br>Participants | MH4 | Summary of Medical Conditions | ICH E3 | SAC |
| 1.12. | All<br>Participants | CM1 | Summary of Concomitant Medications | ICH E3 Note: On-Treatment phase includes both On-Treatment and Post-Treatment concomitant medications. | SAC |
| Exposu | Exposure | | | | |
| 1.13. | Safety | EX1 | Summary of Extent of Exposure to Investigational Product | ICH E3 | SAC |

# 12.11.5. Efficacy Tables

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | Primary Efficacy | | | | |
| 2.1. | Analysis | EFF_T1 | Analysis of Percent Change from Baseline in Leg Press Strength (%) by Visit - Repeated Measure Mixed Model | | Headline<br>Results & SAC |
| 2.2. | Per Protocol | EFF_T1 | Analysis of Percent Change from Baseline in Leg Press Strength (%) by Visit - Repeated Measure Mixed Model | | SAC |
| 2.3. | Analysis | EFF_T1 | Analysis of Change from Baseline in Leg Press Strength (kg) by Visit - Repeated Measure Mixed Model | | SAC |
| 2.4. | Per Protocol | EFF_T1 | Analysis of Change from Baseline in Leg Press Strength (kg) by Visit- Repeated Measure Mixed Model | | SAC |
| 2.5. | Analysis | EFF_T2 | Bayesian Analysis of Percentage Change from Baseline in Leg<br>Press Strength (%) by Visit | | Headline<br>Results & SAC |
| 2.6. | Analysis | EFF_T3 | Descriptive Summary of Change and Percent Change from Baseline in Leg Press Strength by Visit | Summarize the data for change from baseline, percentage change from baseline and ratio to baseline along with the data at each visit for parameters Last Successful Lift 1-Rep Max (kg), Number of Successful Lifts and Starting Lift Weight (kg). | Headline<br>Results & SAC |

| 2.7. | Per Protocol | EFF_T3 | Descriptive Summary of Change and Percent Change from Baseline in Leg Press Strength by Visit | Summarize the data for change from baseline, percentage change from baseline and ratio to baseline along with the data at each visit for parameters Last Successful Lift 1-Rep Max (kg), Number of Successful Lifts and Starting Lift Weight (kg). | SAC |
|---|---|---|---|---|---|
| 2.8. | Analysis | EFF_T1 | Analysis of Percent Change from Baseline in Leg Press Strength (%) by Visit - Repeated Measure Mixed Model with Exploratory Covariate | Add the exploratory covariates predicted FEV1 and BMI at baseline in the same model for Table 2.1. Update the shell footnote by adding the exploratory covariates | SAC |
| Second | ary Efficacy | | | | |
| 2.9. | Analysis | EFF_T1 | Analysis of Change from Baseline in Appendicular (kg), and Total Lean Mass (kg) as Assessed by Dual-energy X-ray Absorptiometry by Visit - Repeated Measure Mixed Model | Similar shell as EFF_T1, add a by line for Parameter under the Sex p-value is not required | Headline<br>Results & SAC |
| 2.10. | Analysis | EFF_T1 | Analysis of Percent Change from Baseline in Appendicular (%), and Total Lean Mass (%) as Assessed by Dual-energy X-ray Absorptiometry by Visit - Repeated Measure Mixed Model | Similar shell as EFF_T1, add a by line for Parameter under the Sex p-value is not required | SAC |
| 2.11. | Analysis | EFF_T3 | Descriptive Summary of Change and Percent Change from Baseline in Appendicular and Total Lean Mass as Assessed by Dual-energy X-ray Absorptiometry by Visit | Summarize the data for change from baseline, percentage change from baseline and ratio to baseline along with the data at each visit | Headline<br>Results & SAC |
| 2.12. | Analysis | EFF_T1 | Analysis of Change from Baseline in PROactive Total Score,<br>Difficulty and Amount Scores by Visit- Repeated Measure Mixed<br>Model | Similar shell as EFF_T1, add a by line for Parameter under the Sex p-value is not required | Headline<br>Results & SAC |

| 2.13. | Per Protocol | EFF_T1 | Analysis of Change from Baseline in PROactive Total Score,<br>Difficulty and Amount Scores by Visit- Repeated Measure Mixed<br>Model | Similar shell as EFF_T1, add a by line for Parameter under the Sex p-value is not required | SAC |
|---|---|---|---|---|---|
| 2.14. | Analysis | EFF_T2 | Bayesian Analysis of Change from Baseline in PROactive Total Score by Visit | | Headline<br>Results & SAC |
| 2.15. | Analysis | EFF_T3 | Descriptive Summary of Change from Baseline in PROactive Total Score, Difficulty and Amount Scores by Visit | Summarize the data for change from baseline and ratio to baseline along with the data at each visit | Headline<br>Results & SAC |
| 2.16. | Per Protocol | EFF_T3 | Descriptive Summary of Change from Baseline in PROactive Total Score, Difficulty and Amounts Scores by Visit | Summarize the data for change from baseline and ratio to baseline along with the data at each visit | SAC |
| 2.17. | Analysis | EFF_T1 | Analysis of Change from Baseline in COPD Assessment Test (CAT) score by Visit- Repeated Measure Mixed Model | Similar shell as EFF_T1, p-value is not required | SAC |
| 2.18. | Analysis | EFF_T6 | Responder Analysis of COPD Assessment Test (CAT) | | SAC |
| 2.19. | Analysis | EFF_T3 | Descriptive Summary of Change from Baseline in COPD<br>Assessment Test (CAT) score by Visit | Summarize the data for change from baseline and ratio to baseline along with the data at each visit | SAC |
| 2.20. | Analysis | EFF_T7 | Analysis of Change from Baseline in St George Respiratory<br>Questionnaire (SGRQ) Total Score and Domains Score at Day<br>90 - ANCOVA Model | | Headline<br>Results & SAC |
| 2.21. | Per Protocol | EFF_T7 | Analysis of Change from Baseline in St George Respiratory<br>Questionnaire (SGRQ) Total Score and Domains Score at Day<br>90 – ANCOVA Model | | SAC |
| 2.22. | Analysis | EFF_T6 | Responder Analysis of St George Respiratory Questionnaire (SGRQ) | | SAC |
| 2.23. | Analysis | EFF_T2 | Bayesian Analysis of Change from Baseline in St George<br>Respiratory Questionnaire (SGRQ) Total Score at Day 90 | Same as EFF_T2, remove the visit column | Headline<br>Results & SAC |

| 2.24. | Analysis | EFF_T3 | Descriptive Summary of Change from Baseline in St George<br>Respiratory Questionnaire (SGRQ) Total Score and Domains<br>Scores by Visit | Summarize the data for change from baseline and ratio to baseline along with the data at each visit | Headline<br>Results & SAC |
|---|---|---|---|---|---|
| 2.25. | Per Protocol | EFF_T3 | Descriptive Summary of Change from Baseline in St George<br>Respiratory Questionnaire (SGRQ) Total Score and Domains<br>Scores by Visit | Summarize the data for change from baseline and ratio to baseline along with the data at each visit | SAC |
| 2.26. | Analysis | EFF_T1 | Analysis of Change from baseline in total Short Physical<br>Performance Battery (SPPB) score and times for chair rise (sec)<br>and 4 m gait speed (sec) by Visit - Repeated Measure Mixed<br>Model | Similar shell as EFF_T1, add a by line for Parameter under the Sex p-value is not required | Headline<br>Results & SAC |
| 2.27. | Per Protocol | EFF_T1 | Analysis of Change from baseline in total Short Physical<br>Performance Battery (SPPB) score and times for chair rise (sec)<br>and 4 m gait speed (sec) by Visit - Repeated Measure Mixed<br>Model | Similar shell as EFF_T1, add a by line for Parameter under the Sex p-value is not required | SAC |
| 2.28. | Analysis | EFF_T2 | Bayesian Analysis of Change from Baseline in Times for chair rise (sec) by Visit | | Headline<br>Results & SAC |
| 2.29. | Analysis | EFF_T3 | Descriptive Summary of Change from baseline in total Short Physical Performance Battery (SPPB) score and times for chair rise and 4 m gait speed by Visit | Summarize the data for change from baseline and ratio to baseline along with the data at each visit | Headline<br>Results & SAC |
| 2.30. | Per Protocol | EFF_T3 | Descriptive Summary of Change from baseline in total Short Physical Performance Battery (SPPB) score and times for chair rise and 4 m gait speed by Visit | Summarize the data for change from baseline and ratio to baseline along with the data at each visit | SAC |
| 2.31. | Analysis | EFF_T7 | Analysis of Change from Baseline in Constant Work Rate (CWR) Duration (sec) from Endurance Shuttle Walking Test at Day 90 – ANCOVA model | Similar shell as EFF_T7, remove the column 'Parameter' | Headline<br>Results & SAC |
| 2.32. | Per Protocol | EFF_T7 | Analysis of Change from Baseline in Constant Work Rate (CWR) Duration (sec) from Endurance Shuttle Walking Test at Day 90 – ANCOVA model | Similar shell as EFF_T7, remove the column 'Parameter' | SAC |

| 2.33. | Analysis | EFF_T7 | Analysis of Percent Change from Baseline in Constant Work Rate (CWR) Duration (%) from Endurance Shuttle Walking Test at Day 90 – ANCOVA model | Similar shell as EFF_T7, remove the column 'Parameter' Update footnote [1] as "[1] Lsmeans of percent change from baseline for each treatment group as well as the difference of Ismeans of percent change from baseline is estimated from ANCOVA model with baseline score as the covariate adjusting for the treatment. In case of violation of the assumptions, the same model is fitted with log of ratio to baseline and replacing the covariate baseline with log baseline." | SAC |
|---|---|---|---|---|---|
| 2.34. | Analysis | EFF_T2 | Bayesian Analysis of Change from Baseline in Constant Work<br>Rate (CWR) Duration (sec) from Endurance Shuttle Walking<br>Test at Day 90 | Same as EFF_T2, remove the visit column | Headline<br>Results & SAC |
| 2.35. | Analysis | EFF_T3 | Descriptive Summary of Change and Percent Change from Baseline in Constant Work Rate (CWR) Duration from Endurance Shuttle Walking Test by Visit | Summarize the data for change from baseline, percentage change from baseline and ratio to baseline along with the data at each visit | Headline<br>Results & SAC |
| 2.36. | Per Protocol | EFF_T3 | Descriptive Summary of Change and Percent Change from Baseline in Constant Work Rate (CWR) Duration from Endurance Shuttle Walking Test by Visit | Summarize the data for change from baseline, percentage change from baseline and ratio to baseline along with the data at each visit | SAC |
| 2.37. | Analysis | EFF_T7 | Analysis of Change from Baseline in Peak Performance from Incremental Shuttle Walking Test at Day 90 – ANCOVA Model | Similar shell as EFF_T7, remove the column 'Parameter' | SAC |

| 2.38. | Analysis | EFF_T7 | Analysis of Percent Change from Baseline in Peak Performance from Incremental Shuttle Walking Test (%) at Day 90 – ANCOVA Model | Similar shell as EFF_T7, remove the column 'Parameter' Update footnote [1] as "[1] Lsmeans of percent change from baseline for each treatment group as well as the difference of Ismeans of percent change from baseline is estimated from ANCOVA model with baseline score as the covariate adjusting for the treatment. In case of violation of the assumptions, the same model is fitted with log of ratio to baseline and replacing the covariate baseline with log baseline." | SAC |
|---|---|---|---|---|---|
| 2.39. | Analysis | EFF_T3 | Descriptive Summary of Change and Percent Change from Baseline in Peak Performance from Incremental Shuttle Walking Test by Visit | Summarize the data for change from baseline, percentage change from baseline and ratio to baseline along with the data at each visit. Update footnote as "Note: When there are multiple pre-dose assessments, the highest non-missing pre-dose assessment from day -9 and day 1 is identified and captured as "Baseline (Derived)" visit" | SAC |
| 2.40. | Analysis | EFF_T3 | Descriptive Summary of Change from Baseline in Physical Activity Measures as Assessed via an Accelerometer. | | SAC |
| 2.41. | Analysis | EFF_T8 | Descriptive Summary of Patient Global Impression of Change | | SAC |
| 2.42. | Analysis | EFF_T10 | Descriptive Summary of Patient Global Rating of Severity. | | SAC |
| 2.43. | Analysis | EFF_T3 | Descriptive Summary of Change from Baseline in FEV1 (L) by Visit | This table will include both FEV1 (L) and Percent Predicted FEV1. | SAC |

| 2.44. | Analysis | EFF_T3 | Descriptive Summary of Change from Baseline in Sniff Nasal Inspiratory Pressure (SnIP) by Visit | | SAC |
|---|---|---|---|---|---|
| Explora | Exploratory | | | | |
| 2.45. | Analysis | EFF_T3 | Descriptive Summary of Change from Baseline in Handgrip strength | First left hand, then right hand | SAC |
| 2.46. | Analysis | EFF_T5 | Descriptive Summary of Change from Baseline in PROactive total and domains scores in different levels of PGIC | | SAC |
| 2.47. | Analysis | EFF_T4 | Analysis of Change from Baseline in Leg Press Strength (kg) by Visit excluding the site PPD (Impact analysis) - Repeated Measure Mixed Model | Fit the model for Table 2.3 by excluding the site PPD. | SAC |

# 12.11.6. Efficacy Figures

| Efficacy: F | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Leg Streng | Leg Strength | | | | |
| 2.1 | Analysis | EFF_F1 | Line Plot of Adjusted Mean (90% CI) Change from Baseline in<br>Leg Press Strength (kg) Over Time – Repeated Measure<br>Mixed Model | Separately for each gender Use the same footnote about model specification as in the corresponding analysis table | SAC |
| 2.2 | Analysis | EFF_F1 | Line Plot of Adjusted Mean (90% CI) Percent Change from Baseline in Leg Press Strength (%) Over Time – Repeated Measure Mixed Model | Separately for each gender Use the same footnote about model specification as in the corresponding analysis table | SAC |
| Lean Mass | | | | | |
| 2.3 | Analysis | EFF_F1 | Line Plot of Adjusted Mean (90% CI) Change from Baseline in<br>Appendicular Lean Mass (kg) and Total Lean Mass (kg) as<br>Assessed by Dual-energy X-ray Absorptiometry Over Time –<br>Repeated Measure Mixed Model | Separately for each gender by parameter Use the same footnote about model specification as in the corresponding analysis table | SAC |
| Functional | Tests | | | | |
| 2.4 | Analysis | EFF_F1 | Line Plot of Adjusted Mean (90% CI) Change from Baseline in PROactive Total Score, Difficulty and Amount Scores Over Time - Repeated Measure Mixed Model | Separately for each gender by parameter Use the same footnote about model specification as in the corresponding analysis table | SAC |
| 2.5 | Analysis | EFF_F1 | Line Plot of Adjusted Mean (90% CI) Change from Baseline in COPD Assessment Test (CAT) score Over Time - Repeated Measure Mixed Model | Separately for each gender Use the same footnote about model specification as in the corresponding analysis table | SAC |

| 2.6 | Analysis | EFF_F1 | Line Plot of Adjusted Mean (90% CI) Change from Baseline in total Short Physical Performance Battery (SPPB) score and times for chair rise (sec) and 4 m gait speed (sec) – Repeated Measure Mixed Model | Separately for each gender by parameter Use the same footnote about model specification as in the corresponding analysis table | SAC |
|---|---|---|---|---|---|
| Exploratory | y Variable | | | | |
| 2.7 | Analysis | LB9 | Box Plot: Change from Baseline in FEV1 (L) | Separately for each gender, X-axis is visit, Y-axis is change from baseline in FEV1 values; | SAC |
| 2.8 | Analysis | LB9 | Box Plot: Change from Baseline in Sniff Nasal Inspiratory Pressure (Snip) | Separately for each gender, X-axis is visit, Y-axis is change from baseline in Snip values; | SAC |
| 2.9 | Analysis | EFF_F1 | Descriptive Mean Change from Baseline in Average Daily Steps over Time | | SAC |

# 12.11.7. Safety Tables

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | Adverse Events (AEs) | | | | |
| 3.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | Headline<br>Results & SAC |
| 3.2. | Safety | AE5A | Summary of Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | For AEs reported more than once by a subject, the most severe intensity will be included. | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.3. | Safety | AE3 | Summary of Common Adverse Events by Overall Frequency | ICH E3 Note: Common adverse event is defined as events occurring more than one in either gender. | SAC |
| 3.4. | Safety | AE3 | Summary of Common Severe Adverse Events by Overall Frequency | ICH E3 Note: Common adverse event is defined as events occurring more than one in either gender. | SAC |
| 3.5. | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term. | ICH E3 | SAC |
| 3.6. | Safety | AE15 | Summary of Common Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT Note: Common adverse event is defined as events occurring more than one in either gender. | SAC |
| 3.7. | Safety | AE3 | Summary of Common Drug-Related Severe Adverse Events by Overall Frequency | ICH E3 Note: Common adverse event is defined as events occurring more than one in either gender. | SAC |
| Serious | and Other Sig | nificant Adverse | Events Events | | |
| 3.8. | Safety | AE3 | Summary of Fatal Serious Adverse Events | | SAC |
| 3.9. | Safety | AE3 | Summary of Drug-Related Fatal Serious Adverse Events | | SAC |
| 3.10. | Safety | AE3 | Summary of Serious Adverse Events by System Organ Class | | SAC |
| 3.11. | Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class | FDAAA, EudraCT | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.12. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | |
| 3.13. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | IDSL | SAC |
| Specia | I Interest AEs | | | | |
| 3.14. | Safety | AE3 | Summary of Adverse Events of Special Interest | IDSL – To display by page for CV events and Liver events | Headline<br>Results & SAC |
| Labora | tory: Chemistr | y | | | |
| 3.15. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit | ICH E3 | SAC |
| 3.16. | Safety | LB16 | Summary of Chemistry Results by Maximum Grade Increases Post-baseline Relative to Baseline | ICH E3 | SAC |
| 3.17. | Safety | LB4 | Summary of Chemistry Shifts from Baseline Relative to Normal Range | IDSL | SAC |
| Labora | tory: Haematol | ogy | | | |
| 3.18. | Safety | LB1 | Summary of Haematology Changes from Baseline | ICH E3 | SAC |
| 3.19. | Safety | LB16 | Summary of Haematology Results by Maximum Grade Increases Post-baseline Relative to Baseline | ICH E3 | SAC |
| 3.20. | Safety | LB4 | Summary of Haematology Shifts from Baseline Relative to Normal Range | IDSL | SAC |
| Labora | tory: Urinalysis | S | | | |
| 3.21. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline | ICH E3 | SAC |
| Safety: | Safety: Tables | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | | |
| 3.22. | Safety | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 Including glucose, protein, blood | SAC | | |
| 3.23. | Safety | LB4 | Summary of Urinalysis Shifts from Baseline Relative to Normal Range | IDSL | SAC | | |
| Laborat | tory: Hepatobil | iary (Liver) | | | | | |
| 3.24. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC | | |
| Laborat | tory: Other | | | | | | |
| 3.25. | Safety | LB1 | Summary of Sex/Reproductive Hormones | Summarize Testosterone, Free Testosterone, Sex hormone-binding globulin (SHBG), Follicle-stimulating hormone (FSH), Luteinizing hormone (LH) and Prostate specific antigen (PSA). | SAC | | |
| 3.26. | Safety | LB1 | Summary of Lipid Panel | | SAC | | |
| 3.27. | Safety | LB1 | Summary of hsCRP, Fibrinogen | | SAC | | |
| ECG | | | | | | | |
| 3.28. | Safety | EG1 | Summary of ECG Findings | IDSL | SAC | | |
| 3.29. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | IDSL | SAC | | |
| 3.30. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC | | |
| 3.31. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | IDSL | SAC | | |
| Vital Sig | gns | | | • | | | |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.32. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |
| 3.33. | Safety | VS7 | Summary of Worst Case Vital Signs Results Relative to Normal Range /Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline | IDSL | SAC |
| Biomar | kers | | | | |
| 3.34. | Safety | LB1 | Summary of Change from Baseline in Bone Biomarkers | | SAC |
| 3.35. | Safety | LB1 | Summary of Change from Baseline in Reproductive Tissue Biomarkers | | SAC |
| COPD E | vents | | | | |
| 3.36. | Safety | SAFE_T1 | Summary of COPD Events | | SAC |

# 12.11.8. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory | | | | |
| 3.1. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT | IDSL | SAC |
| 3.2. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin | IDSL | SAC |
| 3.3. | Safety | EFF_F1 | Line Plot of Change from Baseline in Sex/reproductive Hormones Over Time | Each hormone per page | SAC |
| 3.4. | Safety | EFF_F1 | Line Plot of Change from Baseline in Metabolic factors Over Time | Each factor per page | SAC |

## 12.11.9. Pharmacokinetics Tables

| Pharmacokinetics: Table | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.1 | PK | PK01 | Summary of Plasma Concentration Time data | | SAC |

# 12.11.10. ICH Listings

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | All<br>Participants | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | All<br>Participants | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 4. | All<br>Participants | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| 5. | Enrolled | TA1 / CP_RD1x | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 6. | All<br>Participants | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | All<br>Participants | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| 8. | All<br>Participants | POP_L4 | Listing of Protocol Deviations leading to Exclusion from the Per-<br>Protocol Population | | SAC |
| Popula | tions Analysed | | | | |
| 9. | All<br>Participants | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characterist | ics | | |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 10. | All<br>Participants | DM2 | Listing of Demographic Characteristics | ICH E3 Footnote: Age is imputed when full date of birth is not provided. | SAC |
| 11. | All<br>Participants | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 12. | All<br>Participants | CP_CM3 | Listing of Concomitant Medications | IDSL Note: On-Treatment phase includes both On-Treatment and Post-Treatment concomitant medications. | SAC |
| Expos | ure and Treatme | ent Compliance | | | |
| 13. | All<br>Participants | EX3 | Listing of Investigational Product Exposure Data | ICH E3 | SAC |
| Advers | se Events | | | | |
| 14. | Safety | AE8CPa | Listing of All Adverse Events | ICH E3 | SAC |
| 15. | Safety | AE8 | Listing of Drug-Related Adverse Events | | SAC |
| 16. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| Seriou | s and Other Sig | nificant Adverse l | Events | | |
| 17. | Safety | AE8CPa | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| 18. | Safety | AE8 | Listing of Drug-Related Fatal Serious Adverse Events | | SAC |
| 19. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| 20. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |

| ICH: Lis | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 21. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | • |
| 22. | All<br>Participants | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 23. | All<br>Participants | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL only subjects have such events | SAC |
| 24. | All<br>Participants | LIVER 5 | Listing of Liver Monitoring/Stopping Event Reporting | IDSL only subjects have such events | SAC |
| All Lab | oratory | | | | • |
| 25. | Safety | LB5A | Listing of Clinical Chemistry Laboratory Data | ICH E3 | SAC |
| 26. | Safety | LB5A | Listing of Haematology Laboratory Data | ICH E3 | SAC |
| 27. | Safety | LB14 | Listing of Clinical Chemistry Laboratory Data with Character Results | IDSL | SAC |
| 28. | Safety | LB14 | Listing of Clinical Haematology Data with Character Results | IDSL | SAC |
| 29. | Safety | LB5A | Listing of All Urine Analysis Data | ICH E3 | SAC |
| ECG | | | | | |
| 30. | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |
| 31. | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Findings | IDSL | SAC |
| 32. | Safety | EG3 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| I NO I PONIJISTION I I I I I I I I I I I I I I I I I I | | | | Deliverable<br>[Priority] | |
| Vital Sig | gns | | | | |
| 33. | Safety | VS4 | Listing of All Vital Signs for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |
| 34. | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC |

# 12.11.11. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Study F | Population | | | · | · |
| 35. | Enrolled | POP_L1 | Listing of Subject Recruitment by Country and Site Number | | SAC |
| 36. | Screened | ES9 | Listing of Subject Who were Rescreened | | SAC |
| 37. | All<br>Participants | POP_L2 | Listing of Visit Dates | | SAC |
| 38. | Screened | POP_L3 | Listing of Study Population | | SAC |
| 39. | All<br>Participants | POP_L5 | Listing of Disease Stage and Exacerbation History | | SAC |
| 40. | All<br>Participants | MH2 | Listing of Current and Past Medical Conditions at Baseline | | SAC |
| 41. | All<br>Participants | POP_L6 | Listing of Alcohol History and Tobacco Use/Smoking History | | SAC |
| 42. | All<br>Participants | POP_L7 | Listing of Smoking Status Change during the Study | | SAC |
| 43. | All<br>Participants | POP_L8 | Listing of HIV and Hepatitis Test Results | | SAC |
| 44. | Safety | POP_L9 | Listing of Investigational Product Accountability | | SAC |

| Safety | | | | | |
|---|---|---|---|---|---|
| 45. | Safety | SAFE_L1 | Listing of COPD Exacerbation Log | | SAC |
| 46. | Safety | SAFE_L2 | Listing of Hepatic, Prostate and Cardiac Structure assessed via MRI | | SAC |
| 47. | Safety | SAFE_L3 | Listing of Change from baseline of Lipids and Sex hormones | List the sex hormones Testosterone,<br>Free Testosterone, Sex hormone-<br>binding globulin (SHBG), Follicle-<br>stimulating hormone (FSH), Luteinizing<br>hormone (LH) and Prostate specific<br>antigen (PSA). | SAC |
| Primar | y Efficacy | | | | |
| 48. | Analysis | EFF_L1 | Listing of leg Press Strength (kg) Results | | SAC |
| Second | lary Efficacy | | | | |
| 49. | Analysis | EFF_L2 | Listing of Appendicular (kg), and Total Lean Mass (kg) as Assessed by Dual-energy X-ray Absorptiometry (DXA) | | SAC |
| 50. | Analysis | EFF_L3 | Listing of PROactive Endpoints | Total score, difficulty and amount scores will be displayed | SAC |
| 51. | Analysis | EFF_L4 | Listing of Total Short Physical Performance Battery (SPPB) Score and Times for Chair Rise (sec) and 4 m Gait Speed (sec) Results | | SAC |
| 52. | Analysis | EFF_L5 | Listing of Constant Work Rate (CWR) Duration (sec) from Endurance Shuttle Walking Test | | SAC |
| 53. | Analysis | EFF_L6 | Listing of Peak Performance from Incremental Shuttle Walking Test | | SAC |
| 54. | Analysis | EFF_L7 | Listing of COPD Assessment Test (CAT) | | SAC |
| 55. | Analysis | EFF_L8 | Listing of Patient Global Impression of Change | | SAC |
| 56. | Analysis | EFF_L9 | Listing of Patient Global Rating of Severity | | SAC |

| 57. | Analysis | EFF_L10 | Listing of St George Respiratory Questionnaire (SGRQ) Results | Total score, impact, symptoms and activity domain scores derived by SGRQ-c raw scores | SAC |
|---|---|---|---|---|---|
| 58. | Analysis | EFF_L11 | Listing of Spirometry Results | | SAC |
| 59. | Analysis | EFF_L12 | Listing of Sniff Nasal Inspiratory Pressure (SnIP) | | SAC |
| 60. | Analysis | EFF_L13 | Listing of Physical Activity Measures Assessed via an Accelerometer. | | SAC |
| Explora | atory | | | | |
| 61. | Analysis | EFF_L14 | Listing of Handgrip strength | | SAC |
| Pharma | acokinetics | | | | |
| 62. | PK | PK07 | Listing of Plasma Pharmacokinetic Concentration time data | | SAC |
| Suppo | rtive SAS Listin | g | | | |
| 63. | Analysis | | Supportive SAS Listing for the Analysis of Percent Change from Baseline in Leg Press Strength (%) by Visit - Repeated Measure Mixed Model | | SAC |
| 64. | Per Protocol | | Supportive SAS Listing for Analysis of Percent Change from Baseline in Leg Press Strength (%) by Visit - Repeated Measure Mixed Model | | SAC |
| 65. | Analysis | | Supportive SAS Listing for Analysis of Change from Baseline in Leg Press Strength (kg) by Visit - Repeated Measure Mixed Model | | SAC |
| 66. | Per Protocol | | Supportive SAS Listing for Analysis of Change from Baseline in Leg Press Strength (kg) by Visit- Repeated Measure Mixed Model | | SAC |
| 67. | Analysis | | Supportive SAS Listing for Bayesian Analysis of Percentage Change from Baseline in Leg Press Strength (%) by Visit | | SAC |

| 68. | Analysis | Supportive SAS Listing for Analysis of Percent Change from Baseline in Leg Press Strength (%) by Visit - Repeated Measure Mixed Model with Exploratory Covariates | SAC |
|---|---|---|---|
| 69. | Analysis | Supportive SAS Listing for Analysis of Change from Baseline in Appendicular (kg), and Total Lean Mass (kg) as Assessed by Dual-energy X-ray Absorptiometry by Visit - Repeated Measure Mixed Model | SAC |
| 70. | Analysis | Supportive SAS Listing for Analysis of Percent Change from Baseline in Appendicular (%), and Total Lean Mass (%) as Assessed by Dual-energy X-ray Absorptiometry by Visit - Repeated Measure Mixed Model | SAC |
| 71. | Analysis | Supportive SAS Listing for Analysis of Change from Baseline in PROactive Total Score, Difficulty and Amount Scores by Visit-Repeated Measure Mixed Model | SAC |
| 72. | Per Protocol | Supportive SAS Listing for Analysis of Change from Baseline in PROactive Total Score, Difficulty and Amount Scores by Visit-Repeated Measure Mixed Model | SAC |
| 73. | Analysis | Supportive SAS Listing for Bayesian Analysis of Change from Baseline in PROactive Total Score, Difficulty and Amount Score by Visit | SAC |
| 74. | Analysis | Supportive SAS Listing for Analysis of Change from Baseline in COPD Assessment Test (CAT) score by Visit- Repeated Measure Mixed Model | SAC |
| 75. | Analysis | Supportive SAS Listing for Responder Analysis of COPD Assessment Test (CAT) | SAC |
| 76. | Analysis | Supportive SAS Listing for Analysis of Change from Baseline in St George Respiratory Questionnaire (SGRQ) Total Score and Domains Score at Day 90 - ANCOVA | SAC |

| 77. | Per Protocol | Supportive SAS Listing for Analysis of Change from Baseline in St George Respiratory Questionnaire (SGRQ) Total Score and Domains Score at Day 90 – ANCOVA | SAC |
|---|---|---|---|
| 78. | Analysis | Supportive SAS Listing for Responder Analysis of St George Respiratory Questionnaire (SGRQ) | SAC |
| 79. | Analysis | Supportive SAS Listing for Bayesian Analysis of Change from Baseline in St George Respiratory Questionnaire (SGRQ) Total Score at Day 90 | SAC |
| 80. | Analysis | Supportive SAS Listing for Analysis of Change from baseline in total Short Physical Performance Battery (SPPB) score and times for chair rise (sec) and 4 m gait speed (sec) by Visit - Repeated Measure Mixed Model | SAC |
| 81. | Per Protocol | Supportive SAS Listing for Analysis of Change from baseline in total Short Physical Performance Battery (SPPB) score and times for chair rise (sec) and 4 m gait speed (sec) by Visit - Repeated Measure Mixed Model | SAC |
| 82. | Analysis | Supportive SAS Listing for Bayesian Analysis of Change from Baseline in Times for chair rise (sec) by Visit | SAC |
| 83. | Analysis | Supportive SAS Listing for Analysis of Change from Baseline in Constant Work Rate (CWR) Duration (sec) from Endurance Shuttle Walking Test at Day 90 – ANCOVA model | SAC |
| 84. | Per Protocol | Supportive SAS Listing for Analysis of Change from Baseline in Constant Work Rate (CWR) Duration (sec) from Endurance Shuttle Walking Test at Day 90 – ANCOVA model | SAC |
| 85. | Analysis | Supportive SAS Listing for Analysis of Percent Change from Baseline in Constant Work Rate (CWR) Duration (%) from Endurance Shuttle Walking Test at Day 90 – ANCOVA model | SAC |

| 86. | Analysis | Supportive SAS Listing for Bayesian Analysis of Change from Baseline in Constant Work Rate (CWR) Duration (sec) from Endurance Shuttle Walking Test at Day 90 | SAC |
|---|---|---|---|
| 87. | Analysis | Supportive SAS Listing for Analysis of Change from Baseline in Peak Performance from Incremental Shuttle Walking Test at Day 90 – ANCOVA | SAC |
| 88. | Analysis | Supportive SAS Listing for Analysis of Percent Change from Baseline in Peak Performance from Incremental Shuttle Walking Test (%) at Day 90 - ANCOVA | SAC |
| 89. | Analysis | Supportive SAS Listing for Analysis of Change from Baseline in Leg Press Strength (kg) by Visit excluding the site PPD (Impact analysis) - Repeated Measure Mixed Model | SAC |

200182

## 12.12. Appendix 12: Example Mock Shells for Data Displays

## STUDY POPULATION

## Listings

Example : POP\_L1
Protocol: xxxxxxx
Population: Screened


Sex: Female

| <br>Country | Site Id./ Investigator Name | Unique Subject Id | Randomization<br>Number | Assigned Treatment | Treatment<br>Start Date |
|---|---|---|---|---|---|
| | | xxx | xx | xxx | DDMMMYXXX |
| | | xxx | XX | | DDMMMYXXX |

Programming note: continue with Sex= Male


Example : POP\_L2

Protocol: XXXXXXX

Population: All Participants

Listing xx
Listing of Visit Dates

Country: xxxxx
Centre ID: xxxxxx
Investigator: AAAAAA

| Sex | Unique<br>Subjec<br>Id. | Treatment | Nominal CRF<br>Visit | Visit Start<br>Date | Visit End Date | Analysis Visit | t Study Day |
|---|---|---|---|---|---|---|---|
| F | XXXXX | GSK2881078 | _ | DDMMMYYYY | DDMMMYYYY | Screening | -18 |
| | | | Day 1/Visit 3 | 3 DDWWWXXXX | DDMMMYYYY | Day 1 | 1 |
| | | | Visit 4 | DDMMMYYYY | DDMMMYYYY | Visit 4 | XX |
| | | | Visit 5 | DDMMMYYYY | DDMMMYYYY | Visit 5 | XX |
| | | | Unscheduled | DDMMMYYYY | DDMMMYYYY | Visit 6 | XX |
| | | | | DDMMMYYYY | DDMMMYYYY | Visit 7 | XX |
| | | | • • • | | | | |
| | xxxxx | Placebo | Screening | DDMMMYYYY | DDMMMYYYY | Screening | -29 |
| | | | Day 1 | DDMMMYYYY | DDMMMYYYY | Day 1 | -1 |

<sup>[1]</sup> Analysis Visit is the slotted visits and it is derived by applying the slotting algorithm to Visit Start Date. Programmer's note: repeat for each site within country, then repeat for each country.

200182

Example : POP\_L3
Protocol: XXXXXXX

Population: Screened


Listing xx Listing of Study Populations

Sex: Female
Treatment: None

| Site | Randomized | All | Analysis | Per- | |
|-------------|------------|--------------|----------|----------|--------|
| Id./Invest | Ĺ | Participants | | Protocol | Safety |
| gator | | | | | |
| Id./Investi | Ĺ | | | | |
| gator Name | | | | | |
| xxxxx/xxx | No | No | No | No | No |
| xxxxx/xxx | No | No | No | No | No |
| xxxxx/xxx | No | No | No | No | No |

Sex: Female

| Site | Randomized | All | Analysis | Per- | |
|-------------|------------|--------------|----------|----------|--------|
| Id./Investi | - | Participants | | Protocol | Safety |
| gator | | | | | |
| Id./Investi | - | | | | |
| gator Name | | | | | |
| xxxxx/xxx | Yes | Yes | Yes | Yes | Yes |
| xxxxx/xxx | Yes | Yes | Yes | No | No |
| xxxxx/xxx | Yes | No | No | No | No |

Treatment: Placebo

. .

Programmer's note: Include all analysis populations specified in RAP and give its definition as a footnote.

Example : POP L4

Protocol: xxxxxxx 

Population: All Participants

. . .

Listing xx

Listing of Protocol Deviations Leading to Exclusion from the Per-Protocol Population

Sex: Female

Treatment: GSK2881078

| Inv. | Unique<br>Subj. | Age | Protocol Deviations | Deviation Start<br>Date/<br>Day |
|---|---|---|---|---|
| xxxxx | XXX | XX | xxxxxxxxxxxxxxx | DDMMMYXXX/<br>XXX |
| | xxx | XX | xxxxxxxxxxxxxxxx | DDMMMYXXX/<br>XXX |

89

200182

Example : POP\_L5
Protocol: XXXXXXX

cocol: XXXXXXX Page 1 of x

Population: All Participants

Listing xx

Listing of Disease Stage and Exacerbation History

Sex: Female

| | Disease | Age | Exacerbation History | | | |
|---|---|---|---|---|---|---|
| Site Id./ | Initial | (yrs) | (Number | of Exacerbations | in the last $12$ | Months) |
| Unique<br>Subject<br>Id. | Diag. Date | | Without Corticosteroids and/or Antibiotics | Need<br>Corticosteroids<br>and/or<br>Antibiotics | Required<br>Hospitalised | Period Prior to<br>Visit [1] |
| - | | | 11110122100100 | 11110120100 | | |
| xxx/xxx | DDMMMYYYY | XX | XX | XX | XXXX | XX |
| xxx/xxx | DDMMMYYYY | XX | | | | |
| XXX | DDMMMYYYY | XX | | | | |
| XXX | DDMMMYYYY | XX | | | | |
| XXX | DDMMMYYYY | XX | | | | |

<sup>[1]</sup> Period Prior to Visit is the Evaluation Interval considered while collecting Exacerbation history.

200182

Example : POP\_L6


Population: All Participants

Listing xx

Listing of Alcohol and Tobacco Use/Smoking History

Sex: Female

| Site | Alcohol | | Tobacco Use and Smoking History | | | | | |
|---|---|---|---|---|---|---|---|---|
| Id./Uniq | Assessment | Alcohol | Tobacco | Last Smoke | Smokeless | Number of | Years | Pack |
| ue<br>Subject<br>Id | Date | History/#<br>Unit Per<br>Week | Smoking<br>History | Date | Tobacco<br>Use History | Cigarettes<br>per Day | Smoking<br>Tobacco | Year |
| xxx/xxx | DDMMMYYYY | xx/xx | Smoked | DDMMMYYYY | Current<br>User | xxxx | | xx |
| xxx/xxx | DDMMMYYYY | XX | | | | | | |

200182

Example : POP\_L8

Protocol: YYYYYY

Protocol: XXXXXXXX Page 1 of x

Population: All Participants

Listing xx

Listing of HIV and Hepatitis Test Results

Sex: Female

| Site<br>Id./Uniqu<br>e Subject<br>Id. | Sample Date | Age<br>(yrs) | HIV Test<br>Results/[1] | Hepatitis B Test<br>Result | Hepatitis C Test<br>Result/RBA PCR [2] |
|---|---|---|---|---|---|
| xxx/ | DDMMMYYYY | XX | Negative | Non-Reactive | Non-Reactive |
| XXX | DDMMMYYYY | XX | | Non-Reactive | Reactive |
| xxx/ | DDMMMYYYY | XX | | Non-Reactive | Non-Reactive |
| XXX | DDMMMYYYY | XX | | Non-Reactive | Non-Reactive |
| XXX | DDMMMYYYY | XX | | Non-Reactive | Non-Reactive |

<sup>[1]</sup> only when HIV test is reactive;

<sup>[2]</sup> only when Hepatitis C test is reactive

Example : POP\_L9
Protocol: XXXXXXX

Protocol: XXXXXXX Page 1 of x Population: Safety

Listing xx

Listing of Investigational Product Accountability

Sex: Female

Treatment: GSK2881078

| Site<br>Id. | Unique<br>Subject<br>Id. | Compliance<br>Percentage | Date IP<br>Dispensed/<br>Study Day | Date IP Returned / Study Day | Tablets<br>Dispensed | Tablets<br>Returned | Amoun<br>t<br>Taken | Number<br>of<br>Tables<br>Lost | Container<br>Number |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xx | DDMMMYYYY/<br>xx | DDMMMYYY<br>Y/<br>xx | xx | XX | XX | XX | xxxxx |
| | | | | | XX | XX | XX | XX | xxxxxx |
| | | xx | DDMMMYYYY/<br>xx | DDMMMYYY<br>Y/<br>xx | XX | XX | XX | XX | xxxxxx |
| | | | | | XX | XX | XX | XX | Xxxxxx |

Note: Treatment compliance = 100 \* (Total Amount Taken/ (Actual treatment duration in days\* frequency)).

## **EFFICACY**

## **Tables**

Example : EFF\_T1
Protocol: XXXXXXX

Protocol: XXXXXXX
Population: XXXXXXX


Table xx

\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*

| Visit | | Placebo<br>(N=xxx) | GSK2881078<br>(N=xxx) |
|---|---|---|---|
| Visit X,<br>Day X | n<br>Adjusted Mean [1] (SE)<br>90% C.I. | xxx<br>x.xxx (x.xxx)<br>(x.xxx, x.xxx) | xxx<br>x.xxx (x.xxx)<br>(x.xxx, x.xxx) |
| | GSK2881078 vs. Placebo<br>Difference [2]<br>90% C.I.<br>p-value | | x.xxx<br>(x.xxx, x.xxx)<br>xxx |

<sup>[1]</sup> Estimates were calculated from a repeated measures model including the following covariates: Treatment, Day, Treatment\* Day and baseline xxxxxx, with Day as the repeated factor. In case of violation of the assumptions, the same model is fitted with log of ratio to baseline and replacing the covariate baseline xxxxx with log baseline xxxxx. The correlation matrix for within-subject errors used is unstructured.

[2] GSK2881078-Placebo.

200182

Programming note: Please repeat for Sex: Male.

Programming note: Update the footnotes with the appropriate endpoints and covariate as per RAP.

If data has been log-transformed, then use the following shell:

Protocol: XXXXXXX 

Population: XXXXXX

Table EFF T1

#### \*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*

| Visit | | Placebo<br>(N=xxx) | GSK2881078<br>(N=xxx) |
|---|---|---|---|
| Visit X,<br>Day X | n<br>Model-Adjusted Geometric Mean for<br>Ratio to Baseline (90% CI)[1] | xxx<br>xx.xx (x.xxx, x.xxx) | xxx<br>xx.xx (x.xxx, x.xxx) |
| | Adjusted Treatment Ratio of Geometric Means (90% CI)[2] | | xx.xx (x.xxx, x.xxx) |
| | p-value | | XXXX |

<sup>[1]</sup> Estimates were calculated from a repeated measures model including the following covariates: Treatment, Day, Treatment\* Day and baseline xxxxxx, with Day as the repeated factor. In case of violation of the assumptions, the

200182

same model is fitted with log of ratio to baseline and replacing the covariate baseline xxxxx with log baseline xxxxx. The correlation matrix for within-subject errors used is unstructured.

[2] GSK2881078 ratio to Placebo.

Programming note: Please repeat for Sex: Male.

Programming note: Update the footnotes with the appropriate endpoints and covariate as per RAP.

Example : EFF T2

Protocol: XXXXXXX 

Population: XXXXXXX

#### Table xx

#### 

| Visit | | Placebo<br>(N=xxx) | GSK2881078<br>(N=xxx) |
|---|---|---|---|
| Visit X,<br>Day X | n<br>Posterior Adjusted Mean (SD)[1]<br>90% HPD Credible Interval | xxx<br>x.xxx (x.xxx)<br>(x.xxx, x.xxx) | xxx<br>x.xxx (x.xxx)<br>(x.xxx, x.xxx) |
| | GSK2881078 vs. Placebo<br>Posterior adjusted mean for<br>treatment difference [SD][2]<br>90% HPD Credible Interval | | x.xxx<br>(x.xxx, x.xxx) |
| | Posterior probability treatment difference >=x% | | x.xxx |
| | Posterior probability treatment difference >x% | | x.xxx |
| | Posterior probability treatment difference <x%< td=""><td></td><td>x.xxx</td></x%<> | | x.xxx |

[1] Estimates were calculated from a Bayesian repeated measures model including the following covariates: Treatment, Day, Treatment\* Day and baseline xxxxxx, with Day as the repeated factor.

Female

Male

[2] GSK2881078-Placebo.

Note: HPD - Highest Posterior Density.

Programming note: Please repeat for Sex: Male.

Programming note: Update the footnotes with the appropriate endpoints and covariate as per RAP. Add the

probabilities x% based on the domain.

Example : EFF\_T3
Protocol: XXXX

Protocol: XXXX 

Population: XXXXXX Table XX

#### 

Parameter: xxxxxxxxxxxxxxxxxxxxxxx

| | | Placebo | GSK2881078 | Pla | icebo | GSK2881078 |
|---|---|---|---|---|---|---|
| Visit | Statistics | (N=20) | (N=22) | (N=24) | (N=22) | |
| Baseline | n | xx | xx | хх | XX | |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X | |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | |
| | Median | XX.X | XXX.X | XXX.X | XXX.X | |
| | Min. | XX | XX | XX | XXX | |
| | Max. | XXX | XXX | XXX | XXX | |
| Visit X, Day X | n | XX | XX | XX | xx | |
| | Mean | XXX.X | xxx.x | XXX.X | XXX.X | |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | |
| | Median | XX.X | XXX.X | XXX.X | XXX.X | |
| | Min. | XX | XX | XX | XXX | |
| | Max. | XXX | XXX | XXX | XXX | |

| Change from Baseline at Visit | n | XX | XX | XX | XX |
|-------------------------------|--------|-------|-------|-------|-------|
| X, Day X | Mean | XXX.X | xxx.x | XXX.X | XXX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XXX.X | XXX.X | XXX.X |
| | Min. | XX | XX | XX | XXX |
| | Max. | XXX | xxx | XXX | XXX |

(a) Note: When there are multiple pre-dose assessments, the latest non-missing pre-dose assessment is identified and captured as "Baseline (Derived)" visit.

(b) Note: "Visit X, Day X" is considered as Baseline.

Programming note: Repeat for other visits and summarize its change from baseline, percent change from baseline and ratio to baseline whereever applicable Programming note: If the baseline is a derived visit add the footnote (a) else if it is a single visit add footnote (b)

Example : EFF\_T4
Protocol: XXXXXXX
Population: XXXXXXX


Table xx

Analysis of Change from Baseline in Leg Press Strength (kg) by Visit excluding the site PPD (Impact analysis) - Repeated Measure Mixed Model

| Visit | | Placebo<br>(N=xxx) | GSK2881078<br>(N=xxx) |
|---|---|---|---|
| Visit X,<br>Day X | n<br>n1<br>Adjusted Mean [1] (SE)<br>90% C.I. | xxx<br>xxx<br>x.xxx (x.xxx)<br>(x.xxx, x.xxx) | xxx<br>xxx<br>x.xxx (x.xxx)<br>(x.xxx, x.xxx) |
| | GSK2881078 vs. Placebo<br>Difference [2]<br>90% C.I.<br>p-value | | x.xxx<br>(x.xxx, x.xxx)<br>xxx |

200182

[1] Estimates were calculated from a repeated measures model including the following covariates: Treatment, Day, Treatment\* Day and baseline leg strength with Day as the repeated factor. In case of violation of the assumptions, the same model is fitted with log of ratio to baseline and replacing the covariate baseline leg strength with log baseline leg strength. The correlation matrix for within-subject errors used is unstructured.

[2] GSK2881078-Placebo.

Note: nl indicates the number of analysable subjects excluding the site PPD .

Programming note: Please repeat for Sex: Male.

Programming note: Update the footnotes with the appropriate endpoints and covariate as per RAP.

Example : EFF\_T5

Protocol: xxxxxxx 

Population: Analysis

Table XX

Analysis of Change from Baseline in PROactive total and domains scores in different levels of PGIC

Parameter: XXXXXXXXXXX

| Visit | PGIC Level | Statistics | Males<br>(N=XXX) | Females<br>(N=XXX) | Overall<br>(Males + Females)<br>(N=XXX) |
|---|---|---|---|---|---|
| Visit X, | Much Better | n | XX | XX | Xx |
| Day X | | Mean | xx.xx | xx.xx | XX.XX |
| | | SD | XX.XXX | XX.XXX | XX.XXX |
| | | Median | XX.XX | XX.XX | XX.XX |
| | | Min. | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| | | Max. | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Better | n | XX | XX | Xx |
| | | Mean | XX.XX | XX.XX | XX.XX |
| | | SD | XX.XXX | XX.XXX | XX.XXX |
| | | Median | XX.XX | xx.xx | XX.XX |
| | | Min. | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| | | Max. | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X |

Programming Note: Continue with all PGIC Levels and add levels 'Much Worse and Worse' and 'Better and Much Better'

to the existing levels of PGIC. Repeat for Day 90 and Parameters of PROactive Scores.

Example : EFF\_T6
Protocol: XXXXXXX
Population: Analysis


Table XX

#### 

Sex: Female

| Visit | Treatment | N | Responder Rate $n1/n$ (%) | Odds Ratio (90% C.I.) |
|---|---|---|---|---|
| Visit X, Day | GSK2881078 | XX | xx/xx (xx.x%) | x.xxx (x.xxx, x.xxx) |
| | Placebo | XX | xx/xx (xx.x%) | |

Note: A subject is defined as a responder when the total score at a post-baseline visit decreases

XX or more from baseline total score.

Note: n1 is the number of responders in each treatment group and the percentages are calculated using n

Note: The confidence interval for odds ratio (GSK2881078/Placebo) is calculated using the Exact method. Programming note: continue for the next visit and repeat for Sex: Male.

Example : EFF\_T7
Protocol: XXXXXXX


Population: XXXXXXX

Table XX

#### 

| Parameter | 2 | Placebo<br>(N=xxx) | GSK2881078<br>(N=xxx) |
|---|---|---|---|
| xxxxxxx | n<br>Adjusted Mean [1] (SE)<br>90% C.I. | xxx<br>x.xxx (x.xxx)<br>(x.xxx, x.xxx) | xxx<br>x.xxx (x.xxx)<br>(x.xxx, x.xxx) |
| | GSK2881078 vs. Placebo<br>Difference [2]<br>90% C.I. | | x.xxx<br>(x.xxx, x.xxx) |

<sup>[1]</sup> Lsmeans of change from baseline for each treatment group as well as the difference of lsmeans of change from baseline is estimated from ANCOVA model with baseline score as the covariate adjusting

200182

for the treatment. In case of violation of the assumptions, the same model is fitted with log of ratio to baseline and replacing the covariate baseline with log baseline.
[2] GSK2881078-Placebo.

Example : EFF\_T8
Protocol: XXXXXXXX
Population: Analysis


Table XX

Descriptive Summary of Patient Global Impression of Change

Sex: Female

| Visit | Treatment | N | n | | | | PGIC Categor | У | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Much Worse | Worse | Slightly<br>Worse | No Change | Slightly<br>Better | Better | Much<br>Better |
| Day 14 | GSK2881078<br>Placebo | XX<br>XX | XX | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| Day 28 | GSK2881078<br>Placebo | XX<br>XX | XX<br>XX | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |

Note: The percentages have been calculated based on n.

Programming note: Continue with Visit= Day 56, Day 90 and then repeat for Sex: Male

Example : EFF\_T9

Protocol: XXXXXXXX Page 1 of x

Population: Analysis

Table XX

Descriptive Summary of Patient Global Rating of Severity

Sex: Female

Treatment: Placebo

| Analysis | N | N | N | n | | | PG | RS Category |
|---|---|---|---|---|---|---|---|---|
| Visit | | | None | Mild | Moderate | Severe | Very Severe | |
| Baseline | XX | XX | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | XX | XX | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Day 90 | xx | XX | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | XX | XX | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

... • •

Programming note: repeat for Sex: Male

# **Figures**

Example : EFF\_F1
Protocol: XXXXXXX

Population: XXXXXXXX Figure XX



## Listings

Example : EFF\_L1
Protocol: XXXXXX

: XXXXXXX Page 1 of x

Population: Analysis

Listing XX

Listing of Leg Press Strength (kg) Results

Sex: Female

Treatment: XXXXX

| Site Id/<br>Unique<br>Subject Id | Visit /<br>Analysis<br>Visit | Assessment<br>Date/Day | Parameter | Leg Press Performed? (if no, provide reason) | Assessment<br>Value | Change/Percent<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|
| | Unscheduled /<br>Visit X Day | DDMMMYYYY/1 | Number of<br>Successful<br>Lifts | Yes | xx | xxxx / xxx.x |
| | | | | No | | |
| | | | Starting<br>Lift<br>Weight<br>(Unit) | Yes | xx (xxx) | xxxx / xxx.x |
| | | | Last<br>Successful<br>Lift 1-RM<br>(Unit) | No | | |

Note: Baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.

Programming note: Sorted by treatment, Center, Subject, Visit and continue for SEX: Male Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment Datetime/Day"

Example : EFF\_L2
Protocol: XXXXXX


Population: Analysis

Listing xx

Listing of Appendicular (kg), and Total Lean Mass (kg) as Assessed by Dual-energy X-ray Absorptiometry

(DXA)

Sex: Female

Treatment: XXXXXXXXXXX

| Site Id/<br>Unique<br>Subject<br>Id | Visit /<br>Analysis<br>Visit | Assessment<br>Date/Day | Appendicula | ar Lean Mass | Total Lean Mass | |
|---|---|---|---|---|---|---|
| | | | Assessment<br>(Unit) | Change from<br>Baseline<br>(Unit) | Assessment<br>(Unit) | Change from Baseline (Unit) |
| xxxx/xxxx | Day 1 /<br>Baseline | DDMMMYYYY/1 | xx (xxx) | | xx (xxx) | |
| | Unscheduled<br>/ Visit X<br>Day X | | xx (xxx) | | xx (xxx) | xxxx / xxx.x |

Note: "Visit 3, Day 1" is considered as Baseline.

Programming note: Sorted by treatment, Center, Subject, Visit and continue for SEX: Male Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment Datetime/Day"

Example : EFF\_L3
Protocol: XXXXXX

Population: Analysis


Listing xx Listing of PROactive Endpoints

Sex: Female
Treatment: XXXX

| Site Id/<br>Unique<br>Subject Id | Analysis Visit | Individual Component Score | | Total Score | |
|---|---|---|---|---|---|
| | | Amount<br>/Change from<br>Baseline | Difficulty /Change<br>from Baseline | Assessment | Change from<br>Baseline |
| xxxx/xxxx | Baseline | xx | xx | хх | |
| | Visit X Day X | xx /xxx | xx /xxx | xx | xxxx |

Note: "Visit 3, Day 1" is considered as baseline and is calculated as average of the data collected from the 7-day period after Day -9 device dispense.

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment Datetime/Day"
Programming note: Sorted by treatment, Center, Subject, Visit and continue for SEX: Male

Example : EFF\_L4
Protocol: XXXXXX


Population: Analysis

led /
Visit X
Day X

Listing xx

Listing of Total Short Physical Performance Battery (SPPB) Score and Times for Chair Rise (sec) and 4 m Gait Speed (Sec) Results

Sex: Female
Treatment: XXXX

| Site<br>Id/ | Visit /<br>Analysis | SPPB<br>Perfo | Assessment<br>Date/Day | Balance<br>Tests | Gait S <sub>l</sub> | peed Tests | | | Chair Stand | l Test | SPPB<br>Total |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Unique<br>Subjec<br>t Id | Visit | it rmed? | Total<br>Balance<br>Score | Gait<br>Test<br>Perfo<br>rmed? | Walking<br>Aids | Time for the Fastest Walk (Unit) | 4<br>Meter<br>Walk<br>Test<br>Score | Five<br>Successful<br>Stand Time<br>(unit) | Repeated<br>Chair<br>Test<br>Score | Score | |
| xxxx/x<br>xxx | Baseline | Yes<br>No | DDMMMYYYY/1 | XX | Yes | XXXX | xx(xx) | xx | xx (xxx) | xx (xxx) | xxxx |
| | Unschedu | Yes | | | | | | | | | xxxx |

Note: Baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.

Programming note: Sorted by treatment, Center, Subject, Visit and continue for SEX: Male

200182


Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment Datetime/Day"

Example : EFF\_L5
Protocol: XXXXXX

Population: Analysis

Listing xx

Listing of Constant Work Rate (CWR) Duration (sec) from Endurance Shuttle Walking Test

Sex: Female

| Site Id/<br>Unique<br>Subject<br>Id | Visit /<br>Analysis<br>Visit | Assesment<br>Date/Day | Endurance<br>Time<br>(seconds) | Distance<br>Walked<br>(meters) | Reason for<br>Stopping<br>Test | Endurance<br>Time Change<br>from Baseline |
|---|---|---|---|---|---|---|
| | Day<br>1/Baseline | DDMMMYYYY | XX | XX | XXXXX | |
| | Unscheduled<br>/ Visit X<br>Day X | DDMMMYYYY | xx | xx | xxxxx | xxxx |

200182

Note: "Visit 3, Day 1" is considered as Baseline.

Programming note: Sorted by treatment, Center, Subject, Visit and continue for SEX: Male

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment

Datetime/Day"

Example : EFF\_L6
Protocol: XXXXXX


Population: Analysis

Listing xx

Listing of Peak Performance from Incremental Shuttle Walking Test

Sex: Female

Treatment: XXXXXX

| Site Id/<br>Unique<br>Subject<br>Id | Visit /<br>Analysis<br>Visit | Assesment<br>Date/Day | Maximum<br>Distance Walked<br>(meters) | Speed<br>(km/hr) | Endurance<br>Walking<br>Speed<br>Level | Reason for<br>Stopping<br>Test | Max Walked<br>Distance<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|
| | Day -9<br>Day 1 /<br>Baseline | DDMMMYYYY | xxx | xx | xx | xxxxx<br>Reason for<br>Stopping<br>Test | |
| | Unscheduled<br>/ Visit X<br>Day X | DDMMMYYYY | | | | | |

XXXX

200182

Note: When there are multiple pre-dose assessments, the highest non-missing pre-dose assessment from day -9 and day 1 is identified and captured as "Baseline (Derived)" visit.

Programming note: Sorted by treatment, Center, Subject, Visit and continue for SEX: Male

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment Datetime/Day"

Example : EFF\_L7
Protocol: XXXXXXX


Population: Analysis

Listing xx

Listing of COPD Assessment Test (CAT)

Sex: Female

Treatment: XXXXXX

| | Individual Question Score | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Site<br>Id/<br>Unique<br>Subject | Visit /<br>Analysis<br>Visit | Assesment<br>Date/Day | | | | | | | | | Total<br>Score/Chang |
| Id | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | from Baseline |
| xxxxxx/ | Xx | DDMMMYYYY | Xx | XX | XX | XX | XX | XX | XX | XX | |

XXXXXX

xxxxxx/ DDMMMYYYY

xxxxxx Unscheduled

/ Day xx

Note: 1="Frequency of Cough", 2="Amount of Phlegm in My Chest", 3="Tightness in Chest",

4="Breathless Walking Upstairs", 5="Limited Doing Home Activities", 6="Confident Leaving Home",

7="Sleeping Soundly", 8="Amount of Energy".

Note: "Visit 3, Day 1" is considered as Baseline.

Programming note: Sorted by treatment, Center, Subjects, Visit and continue for SEX: Male

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment

Datetime/Day"

Example : EFF\_L8
Protocol: XXXXXX

Protocol: XXXXXX

Population: Analysis


Listing xx

Listing of Patient Global Impression of Change

Sex: Female

Treatment: XXXXXX

DDMMMYYYY/1 xx

| | | | | | PGIC | Category | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site<br>Id/<br>Unique<br>Subject<br>Id | Assessment<br>Date/Day | Visit /<br>Analysis<br>Visit | Much Worse | Worse | Slightly<br>Worse | No Change | Slightly<br>Better | Better | Much<br>Better |
| | DDMMMYYYY<br>/14 | Visit x<br>/ Visit<br>X Day X | No | No | No | No | Yes | No | No |

Programming note: Sorted by treatment, Center, Subjects, Visit and continue for SEX: Male

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment Datetime/Day"

Example : EFF\_L9
Protocol: XXXXXXX
Population: Analysis


Listing xx
Listing of Patient Global Rating of Severity (PGRS)

Sex: Female
Treatmet: XXXXX

| | | | | | Р | GRS Category | |
|---|---|---|---|---|---|---|---|
| Site Id/<br>Unique<br>Subject Id | Assessment<br>Date/Day | Visit /<br>Analysis<br>Visit | None | Mild | Moderate | Severe | Very Severe |
| Xxxx/xxxx | | Baseline<br>/ Visit<br>X Day X | | | | | Yes |

... **.** 


Programming note: Sorted by treatment, Center, Subjects, Visit and continue for SEX: Male

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment

Datetime/Day"

Example : EFF\_L10 Protocol: XXXXXX

Population: Analysis

Listing xx

Listing of St. George Respiratory Questionnaire (SGRQ) Results

Sex: Female
Treamtment: XXXX

| Site Id/ | Visit / | Assessment | In | ndividual Domain | Score | Total | Score |
|---|---|---|---|---|---|---|---|
| Unique<br>Subject<br>Id | Analysis<br>Visit | Date/Day | Symptoms<br>/Change from<br>Baseline | Activity<br>/Change from<br>Baseline | Impacts/Change<br>from Baseline | Assessment | Change<br>from<br>Baseline |
| xxxx/xxxx | Baseline<br>/ Visit X<br>Day X | DDMMMYYYY/1 | xx | xx | xx | xx | XXXX |
| | Unschedul<br>ed /<br>Visit X | DDMMMYYYY/1 | xx /xxx | xx /xxx | xx /xxx | xx | xxxx |

Day X

Note: "Visit 3, Day 1" is considered as Baseline.

Programming note: Sorted by treatment, Center, Subjects, Visit and continue for SEX: Male

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment

Datetime/Day"

Example : EFF L11 Protocol: XXXXXX Population: Analysis


Listing xx Listing of Spirometry Results

Sex: Female Treatment: XXXXX

| Site Id/<br>Unique<br>Subject<br>Id | Visit /<br>Analysis<br>Visit | Assesment<br>Date/Day | FEV1<br>(L) | Predicted<br>FEV1 (L) | Percent<br>Predicted<br>FEV1 (%) | FVC<br>(L) | Predicted<br>FVC (L) | Percent<br>Predicted<br>FVC (%) | FEV1/FVC |
|---|---|---|---|---|---|---|---|---|---|
| xxxx/xxxx | Screening/<br>Baseline | DDMMMYYYY:hh:mm/-xx | XX | XX | XX | xx | XXXXX | XX | xx.x |
| | Day<br>1/Visit X<br>Day X | DDMMMYYYY:hh:mm/1 | xx | xx | xx | XX | xxxxx | xx | xxx.x |

Note: Baseline value will be the latest pre-dose assessment with a non-missing value, including those from

unscheduled visits.

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment

Datetime/Day"

Programming note: Sorted by treatment, Center, Subjects, Visit and continue for SEX: Male

Example : EFF\_L12
Protocol: XXXXXX
Population: Analysis


Listing xx

Listing of Sniff Nasal Inspiratory Pressure (SNIP)

Sex: Female
Treatment: XXXX

| Site Id/<br>Unique<br>Subject<br>Id | Visit /<br>Analysis<br>Visit | Assesment<br>Datetime/Day | Maximum<br>SnIP | Maximum SnIP<br>Change from<br>Baseline |
|---|---|---|---|---|
| xxxx/xxxx | Screening/<br>Baseline | DDMMMYYYY:hh:mm/-xx | XX.X | |
| | Unscheduled | DDMMMYYYY:hh:mm/1 | xxx.x | |

200182

/ Visit X Day X

Note: Baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.

Programming note: Sorted by treatment, Center, Subjects, Visit and continue for SEX: Male

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment Datetime/Day"

Example : EFF\_L13
Protocol: XXXXXX

Population: Analysis


Listing xx Listing of Handgrip Strength

Sex: Female
Treatment: XXXX

| Site Id/<br>Unique<br>Subject<br>Id | Visit /<br>Analysis<br>Visit | Assessment<br>Date/Day | Left or<br>Right | Performed?<br>(No,reason) | Reading 1 | Reading 2 | Reading 3 | Average of<br>3 Readings |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | Day<br>1/Baseline | DDMMMYYYY<br>/-xx | XX | XX | XX | XX | XXXXX | XX |

200182


Unsheduled DDMMMYYYY xx  $\times$  XX  $\times$  X

Note: Baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.

Programming note: Sorted by treatment, Center, Subjects, Visit and continue for SEX: Male

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment

Datetime/Day"

Example : EFF\_L14
Protocol: XXXXXX

Population: Analysis

Listing xx

Listing of Physical Activity Measures Assessed via an Accelerometer

Sex: Female
Treatment: XXXX

| Site Id/ | Analysis Visit | | | | | |
|---|---|---|---|---|---|---|
| Unique | | Weekly average | Weekly Average | Number of | Weekly | Weekly Average |
| Subject Id | | steps | Wear duration | days with | Average | Moderate/vigorous |
| | | | | wear | Vector | activity duration |
| | | | | duration | magnitude | |

| | | | | more than<br>8 h | unit/wear<br>time | |
|---|---|---|---|---|---|---|
| xxxx/xxxx | Baseline | XX | XX | Xx | xx | |
| | Visit X Day X | xx /xxx | xx /xxx | XX | XX | xxxx |

Note: "Visit 3, Day 1" is considered as baseline and is calculated as average of the data collected from the 7-day period after Day -9 device dispense.

Programming note: Use assessment datetime instead of date if time collected and update the label as "Assessment Datetime/Day"

Programming note: Sorted by treatment, Center, Subject, Visit and continue for SEX: Male

# **SAFETY**

## **Tables**

Example: SAFE\_T1
Protocol: 200182
Population: Safety


## Table xx Summary of COPD Events

| | | Female | | | Male | |
|---|---|---|---|---|---|---|
| motal. | Placebo | GSK2881078 | | Total | Placebo | GSK2881078 |
| Total | (N=xx) | (N=xx) | | (N=xx) | (N=xx) | |
| Number of events in total | x (x%) | x (x%) | х | x (x%) | X | (x%) x |
| Number of exacerbating patients | x (x%) | x (x%) | Х | x (x%) | Х | (x%) x |

# Listings

Example: SAFE\_L1


Population: Safety

Listing xx

Listing of COPD Exacerbation Log

Sex: Female
Treatment: XXXX

| Site<br>Id./ | Onset<br>Date/Day/ | Outcome | Primary<br>Cause | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Unique | Resolution | | (Other, | | | | | | | | |
| Subject<br>Id. | Date | | Specify) | | | | | | | | |

| DDMMMYYYY<br>/xx/DDMMYY | XX<br>YY | Other, xxx | No | No | No | No | No | No | No | XXXX |
|---|---|---|---|---|---|---|---|---|---|---|
| DDMMMYYYY/ | 1 xx | XX | | | | | | | Yes, | |

Note: 1= withdrawn due to the exacerbation, 2=corticosteroids taken for this exacerbation, 3=antibiotics taken for this exacerbation, 4= hospitalized due to this exacerbation, 5=visited the emergency room, 6=intubated for this exacerbation, 7=medication taken for this exacerbation, 8=adverse event reference identifier

Programming note: If medications is taken, show the reference identifier; Sorted by treatment, Center, Subjects and continue for SEX: Male


Example: SAFE\_L2
Protocol: XXXXXX

Population: Safety

Listing xx

Listing of Hepatic, Prostate and Cardiac Structure assessed via MRI

Sex: Female
Treatment: XXXX

| Site Id/<br>Unique<br>Subject<br>Id | Visit /<br>Analysis<br>Visit | Assessment<br>Date/Day | Liver<br>Volume<br>(Unit) | Spleen<br>Volume<br>(Unit) | Prostate<br>Volume<br>(Unit) | Left<br>Ventricular<br>Volume<br>(Unit) | Left<br>Ventricular<br>Ejection<br>Fraction | Left Ventricular End Diastolic Volume Index/ Left Ventricular End Systolic Volume Index |
|---|---|---|---|---|---|---|---|---|
| xxxx/xxxx | Day<br>1/Baseline | DDMMMYYYY<br>/1 | XX | XX | xxxxx | xx | xx.x | XX |
| | Unsheduled<br>/ Visit X<br>Day X | DDMMMYYYY<br>/xx | xx | xx | xxxxx | xx | xxx.x | xx |

Note: "Visit 3, Day 1" is considered as Baseline.

Programming note: Sorted by treatment, Center, Subjects, Visit and continue for SEX: Male

200182

Example : SAFE\_L3


Population: Safety

Listing xx

Listing of Change from baseline of Lipids and Sex hormones

Sex: Female
Treatment: XXXX

| Site Id/<br>Unique<br>Subject<br>Id | Test<br>(Units) | Visit /<br>Analysis<br>Visit | Assesment<br>Datetime/Day | Analysis<br>Value | Change from<br>Baseline |
|---|---|---|---|---|---|
| xxxx/xxxx | PSA | Screening/<br>Baseline | DDMMMYYYY:hh:mm/-xx | XX.X | |
| | | Unscheduled<br>/ Visit X<br>Day X | DDMMMYYYY:hh:mm/1 | xxx.x | xxxx |

Note: The baseline value will be the latest pre-dose assessment between Screening and Day 1 with a non-missing value, including those from unscheduled visits.